CLINICAL TRIAL: NCT02450851
Title: Clinical and Genetic Evaluation of Patients With Undiagnosed Disorders Through the Undiagnosed Diseases Network
Brief Title: Clinical and Genetic Evaluation of Individuals With Undiagnosed Disorders Through the Undiagnosed Diseases Network
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150130; 15-HG-0130
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12-11

CONDITIONS: Genetic Disease
Keywords: Rare Diseases; Undiagnosed Diseases; Natural History
MeSH Terms: conditions — Genetic Diseases, Inborn; Rare Diseases; Undiagnosed Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Undiagnosed disorders: Patients with rare, undiagnosed disorders.

SUMMARY:
Without an explanation for severe and sometimes life-threatening symptoms, patients and their families are left in a state of unknown. Many individuals find themselves being passed from physician to physician, undergoing countless and often repetitive tests in the hopes of finding answers and insight about what the future may hold. This long and arduous journey to find a diagnosis does not end for many patients- the Office of Rare Diseases Research (ORDR) notes that 6% of individuals seeking their assistance have an undiagnosed disorder. In 2008, the National Institutes of Health (NIH) Undiagnosed Diseases Program (UDP) was established with the goal of providing care and answers for these individuals with mysterious conditions who have long eluded diagnosis. The NIH UDP is a joint venture of the NIH ORDR, the National Human Genome Research Institute Intramural Research Program (NHGRI-IRP), and the NIH Clinical Research Center (CRC) (1-3). The goals of the NIH UDP are to: (1) provide answers for patients with undiagnosed diseases; (2) generate new knowledge about disease mechanisms; (3) assess the application of new approaches to phenotyping and the use of genomic technologies; and (4) identify potential therapeutic targets, if possible. To date, the UDP has evaluated 3300 medical records and admitted 750 individuals with rare and undiagnosed conditions to the NIH Clinical Center. The NIH UDP has identified more than 70 rare disease diagnoses and several new conditions. The success of the NIH UDP prompted the NIH Common Fund to support the establishment of a network of medical research centers, the Undiagnosed Diseases Network (UDN), for fiscal years 2013-2020. The clinical sites will perform extensive phenotyping, genetic analyses, and functional studies of potential disease-causing variants. The testing performed on patients involves medically indicated studies intended to help reach a diagnosis, as well as research investigations that include a skin biopsy, blood draws, and DNA analysis. In addition, the UDN will further the goals of the UDP by permitting the sharing of personally identifiable phenotypic and genotypic information within the network. By sharing participant information and encouraging collaboration, the UDN hopes to improve the understanding of rare conditions and advance the diagnostic process and care for individuals with undiagnosed diseases.

DETAILED DESCRIPTION:
Without an explanation for severe and sometimes life-threatening symptoms, patients and their families are left in a state of unknown. Many individuals find themselves being passed from physician to physician, undergoing countless and often repetitive tests in the hopes of finding answers and insight about what the future may hold. This long and arduous journey to find a diagnosis does not end for many patients- the Office of Rare Diseases Research (ORDR) notes that 6% of individuals seeking their assistance have an undiagnosed disorder. In 2008, the National Institutes of Health (NIH) Undiagnosed Diseases Program (UDP) was established with the goal of providing care and answers for these individuals with mysterious conditions who have long eluded diagnosis. The NIH UDP is a joint venture of the NIH ORDR, the National Human Genome Research Institute Intramural Research Program (NHGRI-IRP), and the NIH Clinical Research Center (CRC) (1-3). The goals of the NIH UDP are to: (1) provide answers for patients with undiagnosed diseases; (2) generate new knowledge about disease mechanisms; (3) assess the application of new approaches to phenotyping and the use of genomic technologies; and (4) identify potential therapeutic targets, if possible.1-3 Prior to formation of the Undiagnosed Diseases Network (UDN), the UDP had evaluated 3300 medical records, admitted 750 individuals with rare and undiagnosed conditions to the NIH, and identified more than 70 rare disease diagnoses and several new conditions. The success of the NIH UDP prompted the NIH Common Fund to support the establishment of a network of medical research centers, the UDN, for fiscal years 2013-2022. The clinical sites perform extensive phenotyping, genetic analyses, and functional studies of potential disease-causing variants. The testing performed on patients involves medically indicated studies intended to help reach a diagnosis, as well as research investigations that include a skin biopsy, blood draws, and DNA analysis. In addition, the UDN is furthering the goals of the UDP by permitting the sharing of personally identifiable phenotypic and genotypic information within the network. By sharing participant information and encouraging collaboration, the UDN hopes to improve the understanding of rare conditions and advance the diagnostic process and care for individuals with undiagnosed diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

Ideal participants for tier 2-4 evaluations include individuals with:

* One or more objective findings pertinent to the phenotype for which a case was submitted.
* No diagnosis despite evaluation by specialists who assessed the patient for the objective finding(s).
* Agreement for the storage and sharing of information and biomaterials, in an identified fashion amongst the UDN centers, and in a de-identified fashion to research sites beyond the network.

Participants unable to consent can be enrolled.

EXCLUSION CRITERIA:

Individuals who are unlikely to be assigned to tier 2-4 evaluations include those with:

* Reported symptoms with no relevant objective findings.
* A diagnosis explaining objective findings.
* A diagnosis suggested on record review.
* Unwillingness to share data.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with undiagnosed conditions
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2015-09-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Create an integrated and collaborative research community across multiple clinical sites and between laboratory and clinical investigators prepared to investigate the pathophysiology of these new and rare diseases, the impact of the diagnostic p... | Day 1-5 and followup
  Create an integrated and collaborative research community across multiple clinical sites and between laboratory and clinical investigators prepared to investigate the pathophysiology of these new and rare diseases, the impact of the diagnostic process on patients and families, and share this understanding to identify improved options for optimal patient management.
Facilitate research into the etiology of undiagnosed diseases, by collecting and sharing standardized, high-quality clinical and laboratory data including genotyping, phenotyping, and documentation of environmental exposures | Day 1-5 and followup
  Facilitate research into the etiology of undiagnosed diseases, by collecting and sharing standardized, high-quality clinical and laboratory data including genotyping, phenotyping, and documentation of environmental exposures.
Improve the level of diagnosis and care for patients with undiagnosed diseases through the development of common and site-specific protocols designed by an enlarged community of investigators | Day 1-5 and followup
  Improve the level of diagnosis and care for patients with undiagnosed diseases through the development of common and site-specific protocols designed by an enlarged community of investigators.

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (33):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - HudsonAlpha Institute for Biotechnology, Inc., Huntsville, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Lucile Salter Packard Children's Hospital at Stanford, Stanford, California
  - Stanford University, Stanford, California
  - Leland Stanford Junior University, Stanford, California
  - Stanford Hospital and Clinics, Stanford, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine, Miami, Florida
  - Lurie Children s Hospital, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children s Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Harvard T.H. Chan School of Public Health, Boston, Massachusetts
  - Harvard U Faculty of Medicine, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - New York Genome Center, New York, New York
  - Duke University Health System, Durham, North Carolina
  - University of Oregon, Eugene, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Pacific Northwest National Laboratory, Richland, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Rodan LH, Qi W, Ducker GS, Demirbas D, Laine R, Yang E, Walker MA, Eichler F, Rabinowitz JD, Anselm I, Berry GT; Undiagnosed Diseases Network (UDN). 5,10-methenyltetrahydrofolate synthetase deficiency causes a neurometabolic disorder associated with microcephaly, epilepsy, and cerebral hypomyelination. Mol Genet Metab. 2018 Sep;125(1-2):118-126. doi: 10.1016/j.ymgme.2018.06.006. Epub 2018 Jun 15. PMID 30031689
- [Background] DeBalsi KL, Newman JH, Sommerville LJ, Phillips JA 3rd, Hamid R, Cogan J, Fessel JP, Evans AM, Undiagnosed Diseases Network; Undiagnosed Diseases Network; Kennedy AD. A Case Study of Dysfunctional Nicotinamide Metabolism in a 20-Year-Old Male. Metabolites. 2023 Mar 8;13(3):399. doi: 10.3390/metabo13030399. PMID 36984839
- [Background] Shashi V, Schoch K, Spillmann R, Cope H, Tan QK, Walley N, Pena L, McConkie-Rosell A, Jiang YH, Stong N, Need AC, Goldstein DB; Undiagnosed Diseases Network. A comprehensive iterative approach is highly effective in diagnosing individuals who are exome negative. Genet Med. 2019 Jan;21(1):161-172. doi: 10.1038/s41436-018-0044-2. Epub 2018 Jun 15. PMID 29907797
- [Background] Spillmann RC, Tan QK, Reuter C, Schoch K; Undiagnosed Diseases Network; Kohler J, Bonner D, Zastrow D, Alkelai A, Baugh E, Cope H, Marwaha S, Wheeler MT, Bernstein JA, Shashi V; Undiagnosed Diseases Network. A concurrent dual analysis of genomic data augments diagnoses: Experiences of 2 clinical sites in the Undiagnosed Diseases Network. Genet Med. 2023 Apr;25(4):100353. doi: 10.1016/j.gim.2022.12.001. Epub 2022 Dec 5. PMID 36481303
- [Background] Jangam SV, Briere LC, Jay KL, Andrews JC, Walker MA, Rodan LH, High FA; Undiagnosed Diseases Network; Yamamoto S, Sweetser DA, Wangler MF. A de novo missense variant in EZH1 associated with developmental delay exhibits functional deficits in Drosophila melanogaster. Genetics. 2023 Aug 9;224(4):iyad110. doi: 10.1093/genetics/iyad110. PMID 37314226
- [Background] Briere LC, Walker MA, High FA, Cooper C, Rogers CA, Callahan CJ, Ishimura R, Ichimura Y, Caruso PA, Sharma N, Brokamp E, Koziura ME, Mohammad SS, Dale RC, Riley LG; Undiagnosed Diseases Network; Phillips JA, Komatsu M, Sweetser DA. A description of novel variants and review of phenotypic spectrum in UBA5-related early epileptic encephalopathy. Cold Spring Harb Mol Case Stud. 2021 Jun 11;7(3):a005827. doi: 10.1101/mcs.a005827. Print 2021 Jun. PMID 33811063
- [Background] Huang H, Pan J, Spielberg DR, Hanchard NA, Scott DA, Burrage LC, Dai H, Murdock D, Rosenfeld JA, Mohammad A, Huang T, Lindsey AG, Kim H, Chen J, Ramu A, Morrison SA, Dawson ZD, Hu AZ, Tycksen E, Silverman GA, Baldridge D, Wambach JA; Undiagnosed Diseases Network; Pak SC, Brody SL, Schedl T. A dominant negative variant of RAB5B disrupts maturation of surfactant protein B and surfactant protein C. Proc Natl Acad Sci U S A. 2022 Feb 8;119(6):e2105228119. doi: 10.1073/pnas.2105228119. PMID 35121658
- [Background] Yan YL, Titus T, Desvignes T, BreMiller R, Batzel P, Sydes J, Farnsworth D, Dillon D, Wegner J, Phillips JB, Peirce J, Dowd J; Undiagnosed Diseases Network; Buck CL, Miller A, Westerfield M, Postlethwait JH. A fish with no sex: gonadal and adrenal functions partition between zebrafish NR5A1 co-orthologs. Genetics. 2021 Feb 9;217(2):iyaa030. doi: 10.1093/genetics/iyaa030. PMID 33724412
- [Background] Ganapathi M, Friocourt G, Gueguen N, Friederich MW, Le Gac G, Okur V, Loaec N, Ludwig T, Ka C, Tanji K, Marcorelles P, Theodorou E, Lignelli-Dipple A, Voisset C, Walker MA, Briere LC, Bourhis A, Blondel M, LeDuc C, Hagen J, Cooper C, Muraresku C, Ferec C, Garenne A, Lelez-Soquet S, Rogers CA, Shen Y, Strode DK, Bizargity P, Iglesias A, Goldstein A, High FA, Network UD, Sweetser DA, Ganetzky R, Van Hove JLK, Procaccio V, Le Marechal C, Chung WK. A homozygous splice variant in ATP5PO, disrupts mitochondrial complex V function and causes Leigh syndrome in two unrelated families. J Inherit Metab Dis. 2022 Sep;45(5):996-1012. doi: 10.1002/jimd.12526. Epub 2022 Jul 11. PMID 35621276
- [Background] Gumusderelioglu S, Resch L, Brock T; Undiagnosed Diseases Network; Luxton GWG, Cope H, Tan QK, Hopkins C, Starr DA. A humanized Caenorhabditis elegans model of hereditary spastic paraplegia-associated variants in KLC4. Dis Model Mech. 2023 Aug 1;16(8):dmm050076. doi: 10.1242/dmm.050076. Epub 2023 Aug 29. PMID 37565267
- [Background] Reuter CM, Brimble E, DeFilippo C, Dries AM; Undiagnosed Diseases Network; Enns GM, Ashley EA, Bernstein JA, Fisher PG, Wheeler MT. A New Approach to Rare Diseases of Children: The Undiagnosed Diseases Network. J Pediatr. 2018 May;196:291-297.e2. doi: 10.1016/j.jpeds.2017.12.029. Epub 2018 Jan 11. No abstract available. PMID 29331327
- [Background] Keehan L, Jiang MM, Li X, Marom R, Dai H, Murdock D, Liu P, Hunter JV, Heaney JD, Robak L, Emrick L, Lotze T, Blieden LS; Undiagnosed Diseases Network; Lewis RA, Levin AV, Capasso J, Craigen WJ, Rosenfeld JA, Lee B, Burrage LC. A novel de novo intronic variant in ITPR1 causes Gillespie syndrome. Am J Med Genet A. 2021 Aug;185(8):2315-2324. doi: 10.1002/ajmg.a.62232. Epub 2021 May 5. PMID 33949769
- [Background] Shankar SP, Grimsrud K, Lanoue L, Egense A, Willis B, Horberg J, AlAbdi L, Mayer K, Utkur K, Monaghan KG, Krier J, Stoler J, Alnemer M, Shankar PR, Schaffrath R, Alkuraya FS, Brinkmann U, Eriksson LA, Lloyd K, Rauen KA; Undiagnosed Diseases Network. A novel DPH5-related diphthamide-deficiency syndrome causing embryonic lethality or profound neurodevelopmental disorder. Genet Med. 2022 Jul;24(7):1567-1582. doi: 10.1016/j.gim.2022.03.014. Epub 2022 Apr 28. PMID 35482014
- [Background] Merriweather A, Murdock DR, Rosenfeld JA, Dai H, Ketkar S, Emrick L, Nicholas S, Lewis RA; Undiagnosed Diseases Network; Bacino CA, Scott DA, Lee B, Sutton VR, Potocki L, Burrage LC. A novel, de novo intronic variant in POGZ causes White-Sutton syndrome. Am J Med Genet A. 2022 Jul;188(7):2198-2203. doi: 10.1002/ajmg.a.62747. Epub 2022 Apr 9. PMID 35396900
- [Background] Hom J, Marwaha S, Postolova A, Kittle J, Vasquez R, Davidson J, Kohler J, Dries A, Fernandez-Betancourt L, Majcherska M, Dearlove J, Raghavan S, Vogel H, Bernstein JA, Fisher P, Ashley E, Sampson J, Wheeler M; Undiagnosed Diseases Network. A Patient with Sjogren's Syndrome and Subsequent Diagnosis of Inclusion Body Myositis and Light-Chain Amyloidosis. J Gen Intern Med. 2019 Jun;34(6):1058-1062. doi: 10.1007/s11606-019-04931-w. Epub 2019 Mar 18. PMID 30887439
- [Background] Ferreira CR, Xia ZJ, Clement A, Parry DA, Davids M, Taylan F, Sharma P, Turgeon CT, Blanco-Sanchez B, Ng BG, Logan CV, Wolfe LA, Solomon BD, Cho MT, Douglas G, Carvalho DR, Bratke H, Haug MG, Phillips JB, Wegner J, Tiemeyer M, Aoki K; Undiagnosed Diseases Network; Scottish Genome Partnership; Nordgren A, Hammarsjo A, Duker AL, Rohena L, Hove HB, Ek J, Adams D, Tifft CJ, Onyekweli T, Weixel T, Macnamara E, Radtke K, Powis Z, Earl D, Gabriel M, Russi AHS, Brick L, Kozenko M, Tham E, Raymond KM, Phillips JA 3rd, Tiller GE, Wilson WG, Hamid R, Malicdan MCV, Nishimura G, Grigelioniene G, Jackson A, Westerfield M, Bober MB, Gahl WA, Freeze HH. A Recurrent De Novo Heterozygous COG4 Substitution Leads to Saul-Wilson Syndrome, Disrupted Vesicular Trafficking, and Altered Proteoglycan Glycosylation. Am J Hum Genet. 2018 Oct 4;103(4):553-567. doi: 10.1016/j.ajhg.2018.09.003. PMID 30290151
- [Background] Schoch K, Meng L, Szelinger S, Bearden DR, Stray-Pedersen A, Busk OL, Stong N, Liston E, Cohn RD, Scaglia F, Rosenfeld JA, Tarpinian J, Skraban CM, Deardorff MA, Friedman JN, Akdemir ZC, Walley N, Mikati MA, Kranz PG, Jasien J, McConkie-Rosell A, McDonald M, Wechsler SB, Freemark M, Kansagra S, Freedman S, Bali D, Millan F, Bale S, Nelson SF, Lee H, Dorrani N; UCLA Clinical Genomics Center; Undiagnosed Diseases Network; Goldstein DB, Xiao R, Yang Y, Posey JE, Martinez-Agosto JA, Lupski JR, Wangler MF, Shashi V. A Recurrent De Novo Variant in NACC1 Causes a Syndrome Characterized by Infantile Epilepsy, Cataracts, and Profound Developmental Delay. Am J Hum Genet. 2017 Feb 2;100(2):343-351. doi: 10.1016/j.ajhg.2016.12.013. Epub 2017 Jan 26. PMID 28132692
- [Background] Polovitskaya MM, Barbini C, Martinelli D, Harms FL, Cole FS, Calligari P, Bocchinfuso G, Stella L, Ciolfi A, Niceta M, Rizza T, Shinawi M, Sisco K, Johannsen J, Denecke J, Carrozzo R, Wegner DJ, Kutsche K, Tartaglia M, Jentsch TJ. A Recurrent Gain-of-Function Mutation in CLCN6, Encoding the ClC-6 Cl-/H+-Exchanger, Causes Early-Onset Neurodegeneration. Am J Hum Genet. 2020 Dec 3;107(6):1062-1077. doi: 10.1016/j.ajhg.2020.11.004. Epub 2020 Nov 19. PMID 33217309
- [Background] Bashamboo A, Donohoue PA, Vilain E, Rojo S, Calvel P, Seneviratne SN, Buonocore F, Barseghyan H, Bingham N, Rosenfeld JA, Mulukutla SN, Jain M, Burrage L, Dhar S, Balasubramanyam A, Lee B; Members of UDN; Dumargne MC, Eozenou C, Suntharalingham JP, de Silva K, Lin L, Bignon-Topalovic J, Poulat F, Lagos CF, McElreavey K, Achermann JC. A recurrent p.Arg92Trp variant in steroidogenic factor-1 (NR5A1) can act as a molecular switch in human sex development. Hum Mol Genet. 2016 Aug 15;25(16):3446-3453. doi: 10.1093/hmg/ddw186. Epub 2016 Jul 4. PMID 27378692
- [Background] Dai H, Zhu W, Yuan B, Walley N, Schoch K, Jiang YH, Phillips JA, Jones MS, Liu P, Murdock DR, Burrage LC, Lee B, Rosenfeld JA, Xiao R; Undiagnosed Diseases Network. A recurrent single-exon deletion in TBCK might be under-recognized in patients with infantile hypotonia and psychomotor delay. Hum Mutat. 2022 Dec;43(12):1816-1823. doi: 10.1002/humu.24497. Epub 2022 Nov 6. PMID 36317458
- [Background] Ghosh SG, Scala M, Beetz C, Helman G, Stanley V, Yang X, Breuss MW, Mazaheri N, Selim L, Hadipour F, Pais L, Stutterd CA, Karageorgou V, Begtrup A, Crunk A, Juusola J, Willaert R, Flore LA, Kennelly K, Spencer C, Brown M, Trapane P, Hurst ACE, Lane Rutledge S, Goodloe DH, McDonald MT, Shashi V, Schoch K; Undiagnosed Diseases Network; Tomoum H, Zaitoun R, Hadipour Z, Galehdari H, Pagnamenta AT, Mojarrad M, Sedaghat A, Dias P, Quintas S, Eslahi A, Shariati G, Bauer P, Simons C, Houlden H, Issa MY, Zaki MS, Maroofian R, Gleeson JG. A relatively common homozygous TRAPPC4 splicing variant is associated with an early-infantile neurodegenerative syndrome. Eur J Hum Genet. 2021 Feb;29(2):271-279. doi: 10.1038/s41431-020-00717-5. Epub 2020 Sep 8. PMID 32901138
- [Background] Kyle JE, Stratton KG, Zink EM, Kim YM, Bloodsworth KJ, Monroe ME; Undiagnosed Diseases Network; Waters KM, Webb-Robertson BM, Koeller DM, Metz TO. A resource of lipidomics and metabolomics data from individuals with undiagnosed diseases. Sci Data. 2021 Apr 21;8(1):114. doi: 10.1038/s41597-021-00894-y. PMID 33883556
- [Background] Lino Cardenas CL, Briere LC, Sweetser DA, Lindsay ME, Musolino PL. A seed sequence variant in miR-145-5p causes multisystem smooth muscle dysfunction syndrome. J Clin Invest. 2023 Mar 1;133(5):e166497. doi: 10.1172/JCI166497. No abstract available. PMID 36649075
- [Background] Gu F, Wu A, Gordon MG, Vlahos L, Macnamara S, Burke E, Malicdan MC, Adams DR, Tifft CJ, Toro C, Gahl WA, Markello TC. A suite of automated sequence analyses reduces the number of candidate deleterious variants and reveals a difference between probands and unaffected siblings. Genet Med. 2019 Aug;21(8):1772-1780. doi: 10.1038/s41436-019-0434-0. Epub 2019 Jan 31. PMID 30700791
- [Background] Chao HT, Davids M, Burke E, Pappas JG, Rosenfeld JA, McCarty AJ, Davis T, Wolfe L, Toro C, Tifft C, Xia F, Stong N, Johnson TK, Warr CG; Undiagnosed Diseases Network; Yamamoto S, Adams DR, Markello TC, Gahl WA, Bellen HJ, Wangler MF, Malicdan MCV. A Syndromic Neurodevelopmental Disorder Caused by De Novo Variants in EBF3. Am J Hum Genet. 2017 Jan 5;100(1):128-137. doi: 10.1016/j.ajhg.2016.11.018. Epub 2016 Dec 22. PMID 28017372
- [Background] Paul MS, Michener SL, Pan H, Chan H, Pfliger JM, Rosenfeld JA, Lerma VC, Tran A, Longley MA, Lewis RA, Weisz-Hubshman M, Bekheirnia MR, Bekheirnia N, Massingham L, Zech M, Wagner M, Engels H, Cremer K, Mangold E, Peters S, Trautmann J, Mester JL, Guillen Sacoto MJ, Person R, McDonnell PP, Cohen SR, Lusk L, Cohen ASA, Le Pichon JB, Pastinen T, Zhou D, Engleman K, Racine C, Faivre L, Moutton S, Denomme-Pichon AS, Koh HY, Poduri A, Bolton J, Knopp C, Julia Suh DS, Maier A, Toosi MB, Karimiani EG, Maroofian R, Schaefer GB, Ramakumaran V, Vasudevan P, Prasad C, Osmond M, Schuhmann S, Vasileiou G, Russ-Hall S, Scheffer IE, Carvill GL, Mefford H; Undiagnosed Diseases Network; Bacino CA, Lee BH, Chao HT. A syndromic neurodevelopmental disorder caused by rare variants in PPFIA3. Am J Hum Genet. 2024 Jan 4;111(1):96-118. doi: 10.1016/j.ajhg.2023.12.004. PMID 38181735
- [Background] Zastrow DB, Kohler JN, Bonner D, Reuter CM, Fernandez L, Grove ME, Fisk DG; Undiagnosed Diseases Network; Yang Y, Eng CM, Ward PA, Bick D, Worthey EA, Fisher PG, Ashley EA, Bernstein JA, Wheeler MT. A toolkit for genetics providers in follow-up of patients with non-diagnostic exome sequencing. J Genet Couns. 2019 Apr;28(2):213-228. doi: 10.1002/jgc4.1119. PMID 30964584
- [Background] Spillmann RC, McConkie-Rosell A, Pena L, Jiang YH; Undiagnosed Diseases Network; Schoch K, Walley N, Sanders C, Sullivan J, Hooper SR, Shashi V. A window into living with an undiagnosed disease: illness narratives from the Undiagnosed Diseases Network. Orphanet J Rare Dis. 2017 Apr 17;12(1):71. doi: 10.1186/s13023-017-0623-3. PMID 28416019
- [Background] Xiao C, Koziura M, Cope H, Spillman R, Tan K, Hisama FM, Tifft CJ, Toro C. Adults with lysosomal storage diseases in the undiagnosed diseases network. Mol Genet Genomic Med. 2022 Sep;10(9):e2013. doi: 10.1002/mgg3.2013. Epub 2022 Jul 18. PMID 35848209
- [Background] Schoch K, Tan QK, Stong N, Deak KL, McConkie-Rosell A, McDonald MT; Undiagnosed Diseases Network; Goldstein DB, Jiang YH, Shashi V. Alternative transcripts in variant interpretation: the potential for missed diagnoses and misdiagnoses. Genet Med. 2020 Jul;22(7):1269-1275. doi: 10.1038/s41436-020-0781-x. Epub 2020 May 5. PMID 32366967
- [Background] Ferdinandusse S, McWalter K, Te Brinke H, IJlst L, Mooijer PM, Ruiter JPN, van Lint AEM, Pras-Raves M, Wever E, Millan F, Guillen Sacoto MJ, Begtrup A, Tarnopolsky M, Brady L, Ladda RL, Sell SL, Nowak CB, Douglas J, Tian C, Ulm E, Perlman S, Drack AV, Chong K, Martin N, Brault J, Brokamp E, Toro C, Gahl WA, Macnamara EF, Wolfe L; Undiagnosed Diseases Network; Waisfisz Q, Zwijnenburg PJG, Ziegler A, Barth M, Smith R, Ellingwood S, Gaebler-Spira D, Bakhtiari S, Kruer MC, van Kampen AHC, Wanders RJA, Waterham HR, Cassiman D, Vaz FM. An autosomal dominant neurological disorder caused by de novo variants in FAR1 resulting in uncontrolled synthesis of ether lipids. Genet Med. 2021 Apr;23(4):740-750. doi: 10.1038/s41436-020-01027-3. Epub 2020 Nov 26. PMID 33239752
- [Background] Haghighi A, Krier JB, Toth-Petroczy A, Cassa CA, Frank NY, Carmichael N, Fieg E, Bjonnes A, Mohanty A, Briere LC, Lincoln S, Lucia S, Gupta VA, Soylemez O, Sutti S, Kooshesh K, Qiu H, Fay CJ, Perroni V, Valerius J, Hanna M, Frank A, Ouahed J, Snapper SB, Pantazi A, Chopra SS, Leshchiner I, Stitziel NO, Feldweg A, Mannstadt M, Loscalzo J, Sweetser DA, Liao E, Stoler JM, Nowak CB, Sanchez-Lara PA, Klein OD, Perry H, Patsopoulos NA, Raychaudhuri S, Goessling W, Green RC, Seidman CE, MacRae CA, Sunyaev SR, Maas RL, Vuzman D; Undiagnosed Diseases Network, Brigham and Women's Hospital FaceBase Project, Brigham Genomic Medicine (BGM). An integrated clinical program and crowdsourcing strategy for genomic sequencing and Mendelian disease gene discovery. NPJ Genom Med. 2018 Aug 13;3:21. doi: 10.1038/s41525-018-0060-9. eCollection 2018. PMID 30131872
- [Background] Machol K, Jankovic J, Vijayakumar D, Burrage LC, Jain M, Lewis RA, Fuller GN, Xu M, Penas-Prado M, Gule-Monroe MK, Rosenfeld JA, Chen R, Eng CM, Yang Y, Lee BH, Moretti PM; Undiagnosed Diseases Network; Dhar SU. Atypical Alexander disease with dystonia, retinopathy, and a brain mass mimicking astrocytoma. Neurol Genet. 2018 Jul 20;4(4):e248. doi: 10.1212/NXG.0000000000000248. eCollection 2018 Aug. No abstract available. PMID 30046660
- [Background] Johnston JJ, van der Smagt JJ, Rosenfeld JA, Pagnamenta AT, Alswaid A, Baker EH, Blair E, Borck G, Brinkmann J, Craigen W, Dung VC, Emrick L, Everman DB, van Gassen KL, Gulsuner S, Harr MH, Jain M, Kuechler A, Leppig KA, McDonald-McGinn DM, Can NTB, Peleg A, Roeder ER, Rogers RC, Sagi-Dain L, Sapp JC, Schaffer AA, Schanze D, Stewart H, Taylor JC, Verbeek NE, Walkiewicz MA, Zackai EH, Zweier C; Members of the Undiagnosed Diseases Network; Zenker M, Lee B, Biesecker LG. Autosomal recessive Noonan syndrome associated with biallelic LZTR1 variants. Genet Med. 2018 Oct;20(10):1175-1185. doi: 10.1038/gim.2017.249. Epub 2018 Feb 22. PMID 29469822
- [Background] Young JL, Halley MC, Anguiano B, Fernandez L, Bernstein JA, Wheeler MT, Tabor HK; Undiagnosed Diseases Network Consortium. Beyond race: Recruitment of diverse participants in clinical genomics research for rare disease. Front Genet. 2022 Aug 22;13:949422. doi: 10.3389/fgene.2022.949422. eCollection 2022. PMID 36072659
- [Background] Morimoto M, Bhambhani V, Gazzaz N, Davids M, Sathiyaseelan P, Macnamara EF, Lange J, Lehman A, Zerfas PM, Murphy JL, Acosta MT, Wang C, Alderman E; Undiagnosed Diseases Network; Reichert S, Thurm A, Adams DR, Introne WJ, Gorski SM, Boerkoel CF, Gahl WA, Tifft CJ, Malicdan MCV. Bi-allelic ATG4D variants are associated with a neurodevelopmental disorder characterized by speech and motor impairment. NPJ Genom Med. 2023 Feb 10;8(1):4. doi: 10.1038/s41525-022-00343-8. PMID 36765070
- [Background] Frost FG, Morimoto M, Sharma P, Ruaud L, Belnap N, Calame DG, Uchiyama Y, Matsumoto N, Oud MM, Ferreira EA, Narayanan V, Rangasamy S, Huentelman M, Emrick LT, Sato-Shirai I, Kumada S, Wolf NI, Steinbach PJ, Huang Y; Undiagnosed Diseases Network; Pusey BN, Passemard S, Levy J, Drunat S, Vincent M, Guet A, Agolini E, Novelli A, Digilio MC, Rosenfeld JA, Murphy JL, Lupski JR, Vezina G, Macnamara EF, Adams DR, Acosta MT, Tifft CJ, Gahl WA, Malicdan MCV. Bi-allelic SNAPC4 variants dysregulate global alternative splicing and lead to neuroregression and progressive spastic paraparesis. Am J Hum Genet. 2023 Apr 6;110(4):663-680. doi: 10.1016/j.ajhg.2023.03.001. Epub 2023 Mar 24. PMID 36965478
- [Background] Stephen J, Maddirevula S, Nampoothiri S, Burke JD, Herzog M, Shukla A, Steindl K, Eskin A, Patil SJ, Joset P, Lee H, Garrett LJ, Yokoyama T, Balanda N, Bodine SP, Tolman NJ, Zerfas PM, Zheng A, Ramantani G, Girisha KM, Rivas C, Suresh PV, Elkahloun A, Alsaif HS, Wakil SM, Mahmoud L, Ali R, Prochazkova M; Undiagnosed Diseases Network members; Kulkarni AB, Ben-Omran T, Colak D, Morris HD, Rauch A, Martinez-Agosto JA, Nelson SF, Alkuraya FS, Gahl WA, Malicdan MCV. Bi-allelic TMEM94 Truncating Variants Are Associated with Neurodevelopmental Delay, Congenital Heart Defects, and Distinct Facial Dysmorphism. Am J Hum Genet. 2018 Dec 6;103(6):948-967. doi: 10.1016/j.ajhg.2018.11.001. PMID 30526868
- [Background] Tepe B, Macke EL, Niceta M, Weisz Hubshman M, Kanca O, Schultz-Rogers L, Zarate YA, Schaefer GB, Granadillo De Luque JL, Wegner DJ, Cogne B, Gilbert-Dussardier B, Le Guillou X, Wagner EJ, Pais LS, Neil JE, Mochida GH, Walsh CA, Magal N, Drasinover V, Shohat M, Schwab T, Schmitz C, Clark K, Fine A, Lanpher B, Gavrilova R, Blanc P, Burglen L, Afenjar A, Steel D, Kurian MA, Prabhakar P, Gosswein S, Di Donato N, Bertini ES; Undiagnosed Diseases Network; Wangler MF, Yamamoto S, Tartaglia M, Klee EW, Bellen HJ. Bi-allelic variants in INTS11 are associated with a complex neurological disorder. Am J Hum Genet. 2023 May 4;110(5):774-789. doi: 10.1016/j.ajhg.2023.03.012. Epub 2023 Apr 12. PMID 37054711
- [Background] Kurolap A, Kreuder F, Gonzaga-Jauregui C, Duvdevani MP, Harel T, Tammer L, Xin B, Bakhtiari S, Rice J, van Eyk CL, Gecz J, Mah JK, Atkinson D, Cope H, Sullivan JA, Douek AM, Colquhoun D, Henry J, Wlodkowic D, Parman Y, Candayan A, Kocasoy-Orhan E, Ilivitzki A, Soudry S, Leibu R, Glaser F, Sency V; Undiagnosed Diseases Network; Ast G, Shashi V, Fahey MC, Battaloglu E, Jordanova A, Meiner V, Innes AM, Wang H, Elpeleg O, Kruer MC, Kaslin J, Baris Feldman H. Bi-allelic variants in neuronal cell adhesion molecule cause a neurodevelopmental disorder characterized by developmental delay, hypotonia, neuropathy/spasticity. Am J Hum Genet. 2022 Mar 3;109(3):518-532. doi: 10.1016/j.ajhg.2022.01.004. Epub 2022 Feb 1. PMID 35108495
- [Background] Burrage LC, Reynolds JJ, Baratang NV, Phillips JB, Wegner J, McFarquhar A, Higgs MR, Christiansen AE, Lanza DG, Seavitt JR, Jain M, Li X, Parry DA, Raman V, Chitayat D, Chinn IK, Bertuch AA, Karaviti L, Schlesinger AE, Earl D, Bamshad M, Savarirayan R, Doddapaneni H, Muzny D, Jhangiani SN, Eng CM, Gibbs RA, Bi W, Emrick L, Rosenfeld JA, Postlethwait J, Westerfield M, Dickinson ME, Beaudet AL, Ranza E, Huber C, Cormier-Daire V, Shen W, Mao R, Heaney JD, Orange JS; University of Washington Center for Mendelian Genomics; Undiagnosed Diseases Network; Bertola D, Yamamoto GL, Baratela WAR, Butler MG, Ali A, Adeli M, Cohn DH, Krakow D, Jackson AP, Lees M, Offiah AC, Carlston CM, Carey JC, Stewart GS, Bacino CA, Campeau PM, Lee B. Bi-allelic Variants in TONSL Cause SPONASTRIME Dysplasia and a Spectrum of Skeletal Dysplasia Phenotypes. Am J Hum Genet. 2019 Mar 7;104(3):422-438. doi: 10.1016/j.ajhg.2019.01.007. Epub 2019 Feb 14. PMID 30773277
- [Background] Jeffries L, Mis EK, McWalter K, Donkervoort S, Brodsky NN, Carpier JM, Ji W, Ionita C, Roy B, Morrow JS, Darbinyan A, Iyer K, Aul RB, Banka S, Chao KR, Cobbold L, Cohen S, Custodio HM, Drummond-Borg M, Elmslie F, Finanger E, Hainline BE, Helbig I, Hewson S, Hu Y, Jackson A, Josifova D, Konstantino M, Leach ME, Mak B, McCormick D, McGee E, Nelson S, Nguyen J, Nugent K, Ortega L, Goodkin HP, Roeder E, Roy S, Sapp K, Saade D, Sisodiya SM, Stals K, Towner S, Wilson W; Deciphering Developmental Disorders; Genomics England Research Consortium; Undiagnosed Disease Network; Khokha MK, Bonnemann CG, Lucas CL, Lakhani SA. Biallelic CRELD1 variants cause a multisystem syndrome, including neurodevelopmental phenotypes, cardiac dysrhythmias, and frequent infections. Genet Med. 2024 Feb;26(2):101023. doi: 10.1016/j.gim.2023.101023. Epub 2023 Nov 7. PMID 37947183
- [Background] Schneeberger PE, Kortum F, Korenke GC, Alawi M, Santer R, Woidy M, Buhas D, Fox S, Juusola J, Alfadhel M, Webb BD, Coci EG, Abou Jamra R, Siekmeyer M, Biskup S, Heller C, Maier EM, Javaher-Haghighi P, Bedeschi MF, Ajmone PF, Iascone M, Peeters H, Ballon K, Jaeken J, Rodriguez Alonso A, Palomares-Bralo M, Santos-Simarro F, Meuwissen MEC, Beysen D, Kooy RF, Houlden H, Murphy D, Doosti M, Karimiani EG, Mojarrad M, Maroofian R, Noskova L, Kmoch S, Honzik T, Cope H, Sanchez-Valle A; Undiagnosed Diseases Network; Gelb BD, Kurth I, Hempel M, Kutsche K. Biallelic MADD variants cause a phenotypic spectrum ranging from developmental delay to a multisystem disorder. Brain. 2020 Aug 1;143(8):2437-2453. doi: 10.1093/brain/awaa204. PMID 32761064
- [Background] Olahova M, Yoon WH, Thompson K, Jangam S, Fernandez L, Davidson JM, Kyle JE, Grove ME, Fisk DG, Kohler JN, Holmes M, Dries AM, Huang Y, Zhao C, Contrepois K, Zappala Z, Fresard L, Waggott D, Zink EM, Kim YM, Heyman HM, Stratton KG, Webb-Robertson BM; Undiagnosed Diseases Network; Snyder M, Merker JD, Montgomery SB, Fisher PG, Feichtinger RG, Mayr JA, Hall J, Barbosa IA, Simpson MA, Deshpande C, Waters KM, Koeller DM, Metz TO, Morris AA, Schelley S, Cowan T, Friederich MW, McFarland R, Van Hove JLK, Enns GM, Yamamoto S, Ashley EA, Wangler MF, Taylor RW, Bellen HJ, Bernstein JA, Wheeler MT. Biallelic Mutations in ATP5F1D, which Encodes a Subunit of ATP Synthase, Cause a Metabolic Disorder. Am J Hum Genet. 2018 Mar 1;102(3):494-504. doi: 10.1016/j.ajhg.2018.01.020. Epub 2018 Feb 22. PMID 29478781
- [Background] Shashi V, Schoch K, Ganetzky R, Kranz PG, Sondheimer N, Markert ML, Cope H, Sadeghpour A, Roehrs P, Arbogast T, Muraresku C; Undiagnosed Diseases Network; Tyndall AV, Esser MJ, Woodward KE, Ping-Yee Au B, Parboosingh JS, Lamont RE, Bernier FP, Wright NAM, Benseler SM, Parsons SJ, El-Dairi M, Smith EC, Valdez P, Tennison M, Innes AM, Davis EE. Biallelic variants in ribonuclease inhibitor (RNH1), an inflammasome modulator, are associated with a distinctive subtype of acute, necrotizing encephalopathy. Genet Med. 2023 Sep;25(9):100897. doi: 10.1016/j.gim.2023.100897. Epub 2023 May 13. PMID 37191094
- [Background] Barish S, Barakat TS, Michel BC, Mashtalir N, Phillips JB, Valencia AM, Ugur B, Wegner J, Scott TM, Bostwick B; Undiagnosed Diseases Network; Murdock DR, Dai H, Perenthaler E, Nikoncuk A, van Slegtenhorst M, Brooks AS, Keren B, Nava C, Mignot C, Douglas J, Rodan L, Nowak C, Ellard S, Stals K, Lynch SA, Faoucher M, Lesca G, Edery P, Engleman KL, Zhou D, Thiffault I, Herriges J, Gass J, Louie RJ, Stolerman E, Washington C, Vetrini F, Otsubo A, Pratt VM, Conboy E, Treat K, Shannon N, Camacho J, Wakeling E, Yuan B, Chen CA, Rosenfeld JA, Westerfield M, Wangler M, Yamamoto S, Kadoch C, Scott DA, Bellen HJ. BICRA, a SWI/SNF Complex Member, Is Associated with BAF-Disorder Related Phenotypes in Humans and Model Organisms. Am J Hum Genet. 2020 Dec 3;107(6):1096-1112. doi: 10.1016/j.ajhg.2020.11.003. Epub 2020 Nov 23. PMID 33232675
- [Background] Macnamara EF, Schoch K, Glanton E, Fieg E, Brokamp E; Undiagnosed Diseases Network; Signer R, LeBlanc K, McConkie-Rosell A, Palmer CGS. Cases from the Undiagnosed Diseases Network: The continued value of counseling skills in a new genomic era. J Genet Couns. 2019 Apr;28(2):194-201. doi: 10.1002/jgc4.1091. Epub 2019 Jan 24. PMID 30680851
- [Background] Walley NM, Pena LDM, Hooper SR, Cope H, Jiang YH, McConkie-Rosell A, Sanders C, Schoch K, Spillmann RC, Strong K, McCray AT, Mazur P, Esteves C, LeBlanc K; Undiagnosed Diseases Network; Wise AL, Shashi V. Characteristics of undiagnosed diseases network applicants: implications for referring providers. BMC Health Serv Res. 2018 Aug 22;18(1):652. doi: 10.1186/s12913-018-3458-2. PMID 30134969
- [Background] Beijer D, Kim HJ, Guo L, O'Donovan K, Mademan I, Deconinck T, Van Schil K, Fare CM, Drake LE, Ford AF, Kochanski A, Kabzinska D, Dubuisson N, Van den Bergh P, Voermans NC, Lemmers RJ, van der Maarel SM, Bonner D, Sampson JB, Wheeler MT, Mehrabyan A, Palmer S, De Jonghe P, Shorter J, Taylor JP, Baets J. Characterization of HNRNPA1 mutations defines diversity in pathogenic mechanisms and clinical presentation. JCI Insight. 2021 Jul 22;6(14):e148363. doi: 10.1172/jci.insight.148363. PMID 34291734
- [Background] McConkie-Rosell A, Schoch K, Sullivan J, Spillmann RC, Cope H, Tan QK, Palmer CGS; Undiagnosed Disease Network; Hooper SR, Shashi V. Clinical application of a scale to assess genomic healthcare empowerment (GEmS): Process and illustrative case examples. J Genet Couns. 2022 Feb;31(1):59-70. doi: 10.1002/jgc4.1451. Epub 2021 Jun 11. PMID 34115423
- [Background] Pomerantz DJ, Ferdinandusse S, Cogan J, Cooper DN, Reimschisel T, Robertson A, Bican A, McGregor T, Gauthier J, Millington DS, Andrae JLW, Tschannen MR, Helbling DC, Demos WM, Denis S, Wanders RJA, Newman JN, Hamid R, Phillips JA 3rd; Collaborators of UDN. Clinical heterogeneity of mitochondrial NAD kinase deficiency caused by a NADK2 start loss variant. Am J Med Genet A. 2018 Mar;176(3):692-698. doi: 10.1002/ajmg.a.38602. Epub 2018 Feb 1. PMID 29388319
- [Background] Schoch K, Esteves C, Bican A, Spillmann R, Cope H, McConkie-Rosell A, Walley N, Fernandez L, Kohler JN, Bonner D, Reuter C, Stong N, Mulvihill JJ, Novacic D, Wolfe L, Abdelbaki A, Toro C, Tifft C, Malicdan M, Gahl W, Liu P, Newman J, Goldstein DB, Hom J, Sampson J, Wheeler MT; Undiagnosed Diseases Network; Cogan J, Bernstein JA, Adams DR, McCray AT, Shashi V. Clinical sites of the Undiagnosed Diseases Network: unique contributions to genomic medicine and science. Genet Med. 2021 Feb;23(2):259-271. doi: 10.1038/s41436-020-00984-z. Epub 2020 Oct 23. PMID 33093671
- [Background] Luo X, Rosenfeld JA, Yamamoto S, Harel T, Zuo Z, Hall M, Wierenga KJ, Pastore MT, Bartholomew D, Delgado MR, Rotenberg J, Lewis RA, Emrick L, Bacino CA, Eldomery MK, Coban Akdemir Z, Xia F, Yang Y, Lalani SR, Lotze T, Lupski JR, Lee B, Bellen HJ, Wangler MF; Members of the UDN. Clinically severe CACNA1A alleles affect synaptic function and neurodegeneration differentially. PLoS Genet. 2017 Jul 24;13(7):e1006905. doi: 10.1371/journal.pgen.1006905. eCollection 2017 Jul. PMID 28742085
- [Background] Deisseroth CA, Birgmeier J, Bodle EE, Kohler JN, Matalon DR, Nazarenko Y, Genetti CA, Brownstein CA, Schmitz-Abe K, Schoch K, Cope H, Signer R; Undiagnosed Diseases Network; Martinez-Agosto JA, Shashi V, Beggs AH, Wheeler MT, Bernstein JA, Bejerano G. ClinPhen extracts and prioritizes patient phenotypes directly from medical records to expedite genetic disease diagnosis. Genet Med. 2019 Jul;21(7):1585-1593. doi: 10.1038/s41436-018-0381-1. Epub 2018 Dec 5. PMID 30514889
- [Background] Clement A, Blanco-Sanchez B, Peirce JL, Westerfield M. Cog4 is required for protrusion and extension of the epithelium in the developing semicircular canals. Mech Dev. 2019 Feb;155:1-7. doi: 10.1016/j.mod.2018.09.003. Epub 2018 Oct 1. PMID 30287385
- [Background] Kobren SN, Baldridge D, Velinder M, Krier JB, LeBlanc K, Esteves C, Pusey BN, Zuchner S, Blue E, Lee H, Huang A, Bastarache L, Bican A, Cogan J, Marwaha S, Alkelai A, Murdock DR, Liu P, Wegner DJ, Paul AJ; Undiagnosed Diseases Network; Sunyaev SR, Kohane IS. Commonalities across computational workflows for uncovering explanatory variants in undiagnosed cases. Genet Med. 2021 Jun;23(6):1075-1085. doi: 10.1038/s41436-020-01084-8. Epub 2021 Feb 12. PMID 33580225
- [Background] Miller IM, Yashar BM; Undiagnosed Disease Network; Macnamara EF. Continuing a search for a diagnosis: the impact of adolescence and family dynamics. Orphanet J Rare Dis. 2023 Jan 9;18(1):6. doi: 10.1186/s13023-022-02598-x. PMID 36624503
- [Background] Marom R, Burrage LC, Venditti R, Clement A, Blanco-Sanchez B, Jain M, Scott DA, Rosenfeld JA, Sutton VR, Shinawi M, Mirzaa G, DeVile C, Roberts R, Calder AD, Allgrove J, Grafe I, Lanza DG, Li X, Joeng KS, Lee YC, Song IW, Sliepka JM, Batkovskyte D, Washington M, Dawson BC, Jin Z, Jiang MM, Chen S, Chen Y, Tran AA, Emrick LT, Murdock DR, Hanchard NA, Zapata GE, Mehta NR, Weis MA, Scott AA, Tremp BA, Phillips JB, Wegner J, Taylor-Miller T, Gibbs RA, Muzny DM, Jhangiani SN, Hicks J, Stottmann RW, Dickinson ME, Seavitt JR, Heaney JD, Eyre DR; Undiagnosed Diseases Network; Westerfield M, De Matteis MA, Lee B. COPB2 loss of function causes a coatopathy with osteoporosis and developmental delay. Am J Hum Genet. 2021 Sep 2;108(9):1710-1724. doi: 10.1016/j.ajhg.2021.08.002. Epub 2021 Aug 26. PMID 34450031
- [Background] Brownstein CA, Holm IA, Ramoni R, Goldstein DB; Members of the Undiagnosed Diseases Network. Data sharing in the undiagnosed diseases network. Hum Mutat. 2015 Oct;36(10):985-8. doi: 10.1002/humu.22840. Epub 2015 Aug 27. PMID 26220576
- [Background] Mirzaa GM, Chong JX, Piton A, Popp B, Foss K, Guo H, Harripaul R, Xia K, Scheck J, Aldinger KA, Sajan SA, Tang S, Bonneau D, Beck A, White J, Mahida S, Harris J, Smith-Hicks C, Hoyer J, Zweier C, Reis A, Thiel CT, Jamra RA, Zeid N, Yang A, Farach LS, Walsh L, Payne K, Rohena L, Velinov M, Ziegler A, Schaefer E, Gatinois V, Genevieve D, Simon MEH, Kohler J, Rotenberg J, Wheeler P, Larson A, Ernst ME, Akman CI, Westman R, Blanchet P, Schillaci LA, Vincent-Delorme C, Gripp KW, Mattioli F, Guyader GL, Gerard B, Mathieu-Dramard M, Morin G, Sasanfar R, Ayub M, Vasli N, Yang S, Person R, Monaghan KG, Nickerson DA, van Binsbergen E, Enns GM, Dries AM, Rowe LJ, Tsai ACH, Svihovec S, Friedman J, Agha Z, Qamar R, Rodan LH, Martinez-Agosto J, Ockeloen CW, Vincent M, Sunderland WJ, Bernstein JA; Undiagnosed Diseases Network,; Eichler EE, Vincent JB; University of Washington Center for Mendelian Genomics (UW-CMG),; Bamshad MJ. De novo and inherited variants in ZNF292 underlie a neurodevelopmental disorder with features of autism spectrum disorder. Genet Med. 2020 Mar;22(3):538-546. doi: 10.1038/s41436-019-0693-9. Epub 2019 Nov 14. PMID 31723249
- [Background] Mao D, Reuter CM, Ruzhnikov MRZ, Beck AE, Farrow EG, Emrick LT, Rosenfeld JA, Mackenzie KM, Robak L, Wheeler MT, Burrage LC, Jain M, Liu P, Calame D, Kury S, Sillesen M, Schmitz-Abe K, Tonduti D, Spaccini L, Iascone M, Genetti CA, Koenig MK, Graf M, Tran A, Alejandro M; Undiagnosed Diseases Network; Lee BH, Thiffault I, Agrawal PB, Bernstein JA, Bellen HJ, Chao HT. De novo EIF2AK1 and EIF2AK2 Variants Are Associated with Developmental Delay, Leukoencephalopathy, and Neurologic Decompensation. Am J Hum Genet. 2020 Apr 2;106(4):570-583. doi: 10.1016/j.ajhg.2020.02.016. Epub 2020 Mar 19. PMID 32197074
- [Background] Tokita MJ, Chen CA, Chitayat D, Macnamara E, Rosenfeld JA, Hanchard N, Lewis AM, Brown CW, Marom R, Shao Y, Novacic D, Wolfe L, Wahl C, Tifft CJ, Toro C, Bernstein JA, Hale CL, Silver J, Hudgins L, Ananth A, Hanson-Kahn A, Shuster S; Undiagnosed Diseases Network; Magoulas PL, Patel VN, Zhu W, Chen SM, Jiang Y, Liu P, Eng CM, Batkovskyte D, di Ronza A, Sardiello M, Lee BH, Schaaf CP, Yang Y, Wang X. De Novo Missense Variants in TRAF7 Cause Developmental Delay, Congenital Anomalies, and Dysmorphic Features. Am J Hum Genet. 2018 Jul 5;103(1):154-162. doi: 10.1016/j.ajhg.2018.06.005. Epub 2018 Jun 28. PMID 29961569
- [Background] Kury S, van Woerden GM, Besnard T, Proietti Onori M, Latypova X, Towne MC, Cho MT, Prescott TE, Ploeg MA, Sanders S, Stessman HAF, Pujol A, Distel B, Robak LA, Bernstein JA, Denomme-Pichon AS, Lesca G, Sellars EA, Berg J, Carre W, Busk OL, van Bon BWM, Waugh JL, Deardorff M, Hoganson GE, Bosanko KB, Johnson DS, Dabir T, Holla OL, Sarkar A, Tveten K, de Bellescize J, Braathen GJ, Terhal PA, Grange DK, van Haeringen A, Lam C, Mirzaa G, Burton J, Bhoj EJ, Douglas J, Santani AB, Nesbitt AI, Helbig KL, Andrews MV, Begtrup A, Tang S, van Gassen KLI, Juusola J, Foss K, Enns GM, Moog U, Hinderhofer K, Paramasivam N, Lincoln S, Kusako BH, Lindenbaum P, Charpentier E, Nowak CB, Cherot E, Simonet T, Ruivenkamp CAL, Hahn S, Brownstein CA, Xia F, Schmitt S, Deb W, Bonneau D, Nizon M, Quinquis D, Chelly J, Rudolf G, Sanlaville D, Parent P, Gilbert-Dussardier B, Toutain A, Sutton VR, Thies J, Peart-Vissers LELM, Boisseau P, Vincent M, Grabrucker AM, Dubourg C; Undiagnosed Diseases Network; Tan WH, Verbeek NE, Granzow M, Santen GWE, Shendure J, Isidor B, Pasquier L, Redon R, Yang Y, State MW, Kleefstra T, Cogne B; GEM HUGO; Deciphering Developmental Disorders Study; Petrovski S, Retterer K, Eichler EE, Rosenfeld JA, Agrawal PB, Bezieau S, Odent S, Elgersma Y, Mercier S. De Novo Mutations in Protein Kinase Genes CAMK2A and CAMK2B Cause Intellectual Disability. Am J Hum Genet. 2017 Nov 2;101(5):768-788. doi: 10.1016/j.ajhg.2017.10.003. PMID 29100089
- [Background] Dutta D, Briere LC, Kanca O, Marcogliese PC, Walker MA, High FA, Vanderver A, Krier J, Carmichael N, Callahan C, Taft RJ, Simons C, Helman G, Network UD, Wangler MF, Yamamoto S, Sweetser DA, Bellen HJ. De novo mutations in TOMM70, a receptor of the mitochondrial import translocase, cause neurological impairment. Hum Mol Genet. 2020 Jun 3;29(9):1568-1579. doi: 10.1093/hmg/ddaa081. PMID 32356556
- [Background] Accogli A, Calabretta S, St-Onge J, Boudrahem-Addour N, Dionne-Laporte A, Joset P, Azzarello-Burri S, Rauch A, Krier J, Fieg E, Pallais JC; Undiagnosed Diseases Network; McConkie-Rosell A, McDonald M, Freedman SF, Riviere JB, Lafond-Lapalme J, Simpson BN, Hopkin RJ, Trimouille A, Van-Gils J, Begtrup A, McWalter K, Delphine H, Keren B, Genevieve D, Argilli E, Sherr EH, Severino M, Rouleau GA, Yam PT, Charron F, Srour M. De Novo Pathogenic Variants in N-cadherin Cause a Syndromic Neurodevelopmental Disorder with Corpus Collosum, Axon, Cardiac, Ocular, and Genital Defects. Am J Hum Genet. 2019 Oct 3;105(4):854-868. doi: 10.1016/j.ajhg.2019.09.005. PMID 31585109
- [Background] Weng PL, Majmundar AJ, Khan K, Lim TY, Shril S, Jin G, Musgrove J, Wang M, Ahram DF, Aggarwal VS, Bier LE, Heinzen EL, Onuchic-Whitford AC, Mann N, Buerger F, Schneider R, Deutsch K, Kitzler TM, Klambt V, Kolb A, Mao Y, Moufawad El Achkar C, Mitrotti A, Martino J, Beck BB, Altmuller J, Benz MR, Yano S, Mikati MA, Gunduz T, Cope H, Shashi V; Undiagnosed Diseases Network; Trachtman H, Bodria M, Caridi G, Pisani I, Fiaccadori E, AbuMaziad AS, Martinez-Agosto JA, Yadin O, Zuckerman J, Kim A; UCLA Clinical Genomics Center; John-Kroegel U, Tyndall AV, Parboosingh JS, Innes AM, Bierzynska A, Koziell AB, Muorah M, Saleem MA, Hoefele J, Riedhammer KM, Gharavi AG, Jobanputra V, Pierce-Hoffman E, Seaby EG, O'Donnell-Luria A, Rehm HL, Mane S, D'Agati VD, Pollak MR, Ghiggeri GM, Lifton RP, Goldstein DB, Davis EE, Hildebrandt F, Sanna-Cherchi S. De novo TRIM8 variants impair its protein localization to nuclear bodies and cause developmental delay, epilepsy, and focal segmental glomerulosclerosis. Am J Hum Genet. 2021 Feb 4;108(2):357-367. doi: 10.1016/j.ajhg.2021.01.008. Epub 2021 Jan 27. PMID 33508234
- [Background] Shashi V, Pena LD, Kim K, Burton B, Hempel M, Schoch K, Walkiewicz M, McLaughlin HM, Cho M, Stong N, Hickey SE, Shuss CM; Undiagnosed Diseases Network; Freemark MS, Bellet JS, Keels MA, Bonner MJ, El-Dairi M, Butler M, Kranz PG, Stumpel CT, Klinkenberg S, Oberndorff K, Alawi M, Santer R, Petrovski S, Kuismin O, Korpi-Heikkila S, Pietilainen O, Aarno P, Kurki MI, Hoischen A, Need AC, Goldstein DB, Kortum F. De Novo Truncating Variants in ASXL2 Are Associated with a Unique and Recognizable Clinical Phenotype. Am J Hum Genet. 2016 Oct 6;99(4):991-999. doi: 10.1016/j.ajhg.2016.08.017. Epub 2016 Sep 29. PMID 27693232
- [Background] Royer-Bertrand B, Jequier Gygax M, Cisarova K, Rosenfeld JA, Bassetti JA, Moldovan O, O'Heir E, Burrage LC, Allen J, Emrick LT, Eastman E, Kumps C, Abbas S, Van Winckel G; Undiagnosed Diseases Network; Chabane N, Zackai EH, Lebon S, Keena B, Bhoj EJ, Umair M, Li D, Donald KA, Superti-Furga A. De novo variants in CACNA1E found in patients with intellectual disability, developmental regression and social cognition deficit but no seizures. Mol Autism. 2021 Oct 26;12(1):69. doi: 10.1186/s13229-021-00473-3. PMID 34702355
- [Background] Chung HL, Mao X, Wang H, Park YJ, Marcogliese PC, Rosenfeld JA, Burrage LC, Liu P, Murdock DR, Yamamoto S, Wangler MF; Undiagnosed Diseases Network; Chao HT, Long H, Feng L, Bacino CA, Bellen HJ, Xiao B. De Novo Variants in CDK19 Are Associated with a Syndrome Involving Intellectual Disability and Epileptic Encephalopathy. Am J Hum Genet. 2020 May 7;106(5):717-725. doi: 10.1016/j.ajhg.2020.04.001. Epub 2020 Apr 23. PMID 32330417
- [Background] Ma M, Zheng Y, Deng M, Lu S, Pan X, Luo X, Etoundi M, Li-Kroeger D, Worley KC, Burrage LC, Blieden LS, Allworth A, Chen WL, Merla G, Mandriani B, Otten CE, Blanc P, Rosenfeld JA, Dutta D, Yamamoto S, Wangler MF; Undiagnosed Diseases Network; Glass IA, Chen J, Blue E, Prontera P, Rosain J, Marlin S, Lalani SR, Bellen HJ. Heterozygous variants in PLCG1 affect hearing, vision, cardiac, and immune function. medRxiv [Preprint]. 2025 May 29:2024.01.08.23300523. doi: 10.1101/2024.01.08.23300523. PMID 38260438
- [Background] Guillen Sacoto MJ, Tchasovnikarova IA, Torti E, Forster C, Andrew EH, Anselm I, Baranano KW, Briere LC, Cohen JS, Craigen WJ, Cytrynbaum C, Ekhilevitch N, Elrick MJ, Fatemi A, Fraser JL, Gallagher RC, Guerin A, Haynes D, High FA, Inglese CN, Kiss C, Koenig MK, Krier J, Lindstrom K, Marble M, Meddaugh H, Moran ES, Morel CF, Mu W, Muller EA 2nd, Nance J, Natowicz MR, Numis AL, Ostrem B, Pappas J, Stafstrom CE, Streff H, Sweetser DA, Szybowska M; Undiagnosed Diseases Network; Walker MA, Wang W, Weiss K, Weksberg R, Wheeler PG, Yoon G, Kingston RE, Juusola J. De Novo Variants in the ATPase Module of MORC2 Cause a Neurodevelopmental Disorder with Growth Retardation and Variable Craniofacial Dysmorphism. Am J Hum Genet. 2020 Aug 6;107(2):352-363. doi: 10.1016/j.ajhg.2020.06.013. Epub 2020 Jul 20. PMID 32693025
- [Background] Kanca O, Andrews JC, Lee PT, Patel C, Braddock SR, Slavotinek AM, Cohen JS, Gubbels CS, Aldinger KA, Williams J, Indaram M, Fatemi A, Yu TW, Agrawal PB, Vezina G, Simons C, Crawford J, Lau CC; Undiagnosed Diseases Network; Chung WK, Markello TC, Dobyns WB, Adams DR, Gahl WA, Wangler MF, Yamamoto S, Bellen HJ, Malicdan MCV. De Novo Variants in WDR37 Are Associated with Epilepsy, Colobomas, Dysmorphism, Developmental Delay, Intellectual Disability, and Cerebellar Hypoplasia. Am J Hum Genet. 2019 Aug 1;105(2):413-424. doi: 10.1016/j.ajhg.2019.06.014. Epub 2019 Jul 18. PMID 31327508
- [Background] Ferreira CR, Zein WM, Huryn LA, Merker A, Berger SI, Wilson WG, Tiller GE, Wolfe LA, Merideth M, Carvalho DR, Duker AL, Bratke H, Haug MG, Rohena L, Hove HB, Xia ZJ, Ng BG, Freeze HH, Gabriel M, Russi AHS, Brick L, Kozenko M, Earl DL, Tham E, Nishimura G, Phillips JA 3rd, Gahl WA, Hamid R, Jackson AP, Grigelioniene G, Bober MB. Defining the clinical phenotype of Saul-Wilson syndrome. Genet Med. 2020 May;22(5):857-866. doi: 10.1038/s41436-019-0737-1. Epub 2020 Jan 17. PMID 31949312
- [Background] Cope H, Barseghyan H, Bhattacharya S, Fu Y, Hoppman N, Marcou C, Walley N, Rehder C, Deak K, Alkelai A; Undiagnosed Diseases Network; Vilain E, Shashi V. Detection of a mosaic CDKL5 deletion and inversion by optical genome mapping ends an exhaustive diagnostic odyssey. Mol Genet Genomic Med. 2021 Jul;9(7):e1665. doi: 10.1002/mgg3.1665. Epub 2021 May 6. PMID 33955715
- [Background] Grove ME, White S, Fisk DG, Rego S, Dagan-Rosenfeld O, Kohler JN, Reuter CM, Bonner D; Undiagnosed Diseases Network; Wheeler MT, Bernstein JA, Ormond KE, Hanson-Kahn AK. Developing a genomics rotation: Practical training around variant interpretation for genetic counseling students. J Genet Couns. 2019 Apr;28(2):466-476. doi: 10.1002/jgc4.1094. Epub 2019 Feb 1. PMID 30706981
- [Background] LaFlamme CW, Rastin C, Sengupta S, Pennington HE, Russ-Hall SJ, Schneider AL, Bonkowski ES, Almanza Fuerte EP, Galey M, Goffena J, Gibson SB, Allan TJ, Nyaga DM, Lieffering N, Hebbar M, Walker EV, Darnell D, Olsen SR, Kolekar P, Djekidel N, Rosikiewicz W, McConkey H, Kerkhof J, Levy MA, Relator R, Lev D, Lerman-Sagie T, Park KL, Alders M, Cappuccio G, Chatron N, Demain L, Genevieve D, Lesca G, Roscioli T, Sanlaville D, Tedder ML, Hubshman MW, Ketkar S, Dai H, Worley KC, Rosenfeld JA, Chao HT; Undiagnosed Diseases Network; Neale G, Carvill GL; University of Washington Center for Rare Disease Research; Wang Z, Berkovic SF, Sadleir LG, Miller DE, Scheffer IE, Sadikovic B, Mefford HC. Diagnostic Utility of Genome-wide DNA Methylation Analysis in Genetically Unsolved Developmental and Epileptic Encephalopathies and Refinement of a CHD2 Episignature. medRxiv [Preprint]. 2023 Oct 12:2023.10.11.23296741. doi: 10.1101/2023.10.11.23296741. PMID 37873138
- [Background] Lee H, Huang AY, Wang LK, Yoon AJ, Renteria G, Eskin A, Signer RH, Dorrani N, Nieves-Rodriguez S, Wan J, Douine ED, Woods JD, Dell'Angelica EC, Fogel BL, Martin MG, Butte MJ, Parker NH, Wang RT, Shieh PB, Wong DA, Gallant N, Singh KE, Tavyev Asher YJ, Sinsheimer JS, Krakow D, Loo SK, Allard P, Papp JC; Undiagnosed Diseases Network; Palmer CGS, Martinez-Agosto JA, Nelson SF. Diagnostic utility of transcriptome sequencing for rare Mendelian diseases. Genet Med. 2020 Mar;22(3):490-499. doi: 10.1038/s41436-019-0672-1. Epub 2019 Oct 14. PMID 31607746
- [Background] Granadillo JL, Wegner DJ, Paul AJ, Willing M, Sisco K, Tedder ML, Sadikovic B, Wambach JA, Baldridge D, Cole FS; Undiagnosed Diseases Network. Discovery of a novel CHD7 CHARGE syndrome variant by integrated omics analyses. Am J Med Genet A. 2021 Feb;185(2):544-548. doi: 10.1002/ajmg.a.61962. Epub 2020 Nov 13. PMID 33184947
- [Background] Runge K, Mathieu R, Bugeon S, Lafi S, Beurrier C, Sahu S, Schaller F, Loubat A, Herault L, Gaillard S, Pallesi-Pocachard E, Montheil A, Bosio A, Rosenfeld JA, Hudson E, Lindstrom K, Mercimek-Andrews S, Jeffries L, van Haeringen A, Vanakker O, Van Hecke A, Amrom D, Kury S, Ratner C, Jethva R, Gamble C, Jacq B, Fasano L, Santpere G, Lorente-Galdos B, Sestan N, Gelot A, Giacuzz S, Goebbels S, Represa A, Cardoso C, Cremer H, de Chevigny A. Correction: Disruption of NEUROD2 causes a neurodevelopmental syndrome with autistic features via cell-autonomous defects in forebrain glutamatergic neurons. Mol Psychiatry. 2021 Dec;26(12):7852. doi: 10.1038/s41380-021-01234-7. No abstract available. PMID 34282265
- [Background] Deuitch NT, Beckman E, Halley MC, Young JL, Reuter CM, Kohler J, Bernstein JA, Wheeler MT; Undiagnosed Diseases Network; Ormond KE, Tabor HK. "Doctors can read about it, they can know about it, but they've never lived with it": How parents use social media throughout the diagnostic odyssey. J Genet Couns. 2021 Dec;30(6):1707-1718. doi: 10.1002/jgc4.1438. Epub 2021 Jun 6. PMID 34096130
- [Background] Marom R, Zhang B, Washington ME, Song IW, Burrage LC, Rossi VC, Berrier AS, Lindsey A, Lesinski J, Nonet ML, Chen J, Baldridge D, Silverman GA, Sutton VR, Rosenfeld JA, Tran AA, Hicks MJ, Murdock DR, Dai H, Weis M, Jhangiani SN, Muzny DM, Gibbs RA, Caswell R, Pottinger C, Cilliers D, Stals K; Undiagnosed Diseases Network; Eyre D, Krakow D, Schedl T, Pak SC, Lee BH. Dominant negative variants in KIF5B cause osteogenesis imperfecta via down regulation of mTOR signaling. PLoS Genet. 2023 Nov 7;19(11):e1011005. doi: 10.1371/journal.pgen.1011005. eCollection 2023 Nov. PMID 37934770
- [Background] Beziat V, Tavernier SJ, Chen YH, Ma CS, Materna M, Laurence A, Staal J, Aschenbrenner D, Roels L, Worley L, Claes K, Gartner L, Kohn LA, De Bruyne M, Schmitz-Abe K, Charbonnier LM, Keles S, Nammour J, Vladikine N, Maglorius Renkilaraj MRL, Seeleuthner Y, Migaud M, Rosain J, Jeljeli M, Boisson B, Van Braeckel E, Rosenfeld JA, Dai H, Burrage LC, Murdock DR, Lambrecht BN, Avettand-Fenoel V, Vogel TP; Undiagnosed Diseases Network; Esther CR, Haskologlu S, Dogu F, Ciznar P, Boutboul D, Ouachee-Chardin M, Amourette J, Lebras MN, Gauvain C, Tcherakian C, Ikinciogullari A, Beyaert R, Abel L, Milner JD, Grimbacher B, Couderc LJ, Butte MJ, Freeman AF, Catherinot E, Fieschi C, Chatila TA, Tangye SG, Uhlig HH, Haerynck F, Casanova JL, Puel A. Dominant-negative mutations in human IL6ST underlie hyper-IgE syndrome. J Exp Med. 2020 Jun 1;217(6):e20191804. doi: 10.1084/jem.20191804. PMID 32207811
- [Background] Pujol-Gimenez J, Mirzaa G, Blue EE, Albano G, Miller DE, Allworth A, Bennett JT, Byers PH, Chanprasert S, Chen J, Doherty D, Folta AB, Gillentine MA, Glass I, Hing A, Horike-Pyne M, Leppig KA, Parhin A, Ranchalis J, Raskind WH, Rosenthal EA, Schwarze U, Sheppeard S, Strohbehn S, Sybert VP, Timms A, Wener M; University of Washington Center for Mendelian Genomics (UW-CMG)a, Undiagnosed Diseases Network (UDN); Bamshad MJ, Hisama FM, Jarvik GP, Dipple KM, Hediger MA, Stergachis AB. Dominant-negative variant in SLC1A4 causes an autosomal dominant epilepsy syndrome. Ann Clin Transl Neurol. 2023 Jun;10(6):1046-1053. doi: 10.1002/acn3.51786. Epub 2023 May 16. PMID 37194416
- [Background] Meissner LE, Macnamara EF, D'Souza P, Yang J, Vezina G; Undiagnosed Diseases Network; Ferreira CR, Zein WM, Tifft CJ, Adams DR. DYRK1A pathogenic variants in two patients with syndromic intellectual disability and a review of the literature. Mol Genet Genomic Med. 2020 Dec;8(12):e1544. doi: 10.1002/mgg3.1544. Epub 2020 Nov 7. PMID 33159716
- [Background] Johnstone DL, Nguyen TTM, Zambonin J, Kernohan KD, St-Denis A, Baratang NV, Hartley T, Geraghty MT, Richer J, Majewski J, Bareke E, Guerin A, Pendziwiat M, Pena LDM, Braakman HMH, Gripp KW, Edmondson AC, He M, Spillmann RC, Eklund EA, Bayat A, McMillan HJ, Boycott KM, Campeau PM. Early infantile epileptic encephalopathy due to biallelic pathogenic variants in PIGQ: Report of seven new subjects and review of the literature. J Inherit Metab Dis. 2020 Nov;43(6):1321-1332. doi: 10.1002/jimd.12278. Epub 2020 Aug 3. PMID 32588908
- [Background] Splinter K, Adams DR, Bacino CA, Bellen HJ, Bernstein JA, Cheatle-Jarvela AM, Eng CM, Esteves C, Gahl WA, Hamid R, Jacob HJ, Kikani B, Koeller DM, Kohane IS, Lee BH, Loscalzo J, Luo X, McCray AT, Metz TO, Mulvihill JJ, Nelson SF, Palmer CGS, Phillips JA 3rd, Pick L, Postlethwait JH, Reuter C, Shashi V, Sweetser DA, Tifft CJ, Walley NM, Wangler MF, Westerfield M, Wheeler MT, Wise AL, Worthey EA, Yamamoto S, Ashley EA; Undiagnosed Diseases Network. Effect of Genetic Diagnosis on Patients with Previously Undiagnosed Disease. N Engl J Med. 2018 Nov 29;379(22):2131-2139. doi: 10.1056/NEJMoa1714458. Epub 2018 Oct 10. PMID 30304647
- [Background] Boonsawat P, Joset P, Steindl K, Oneda B, Gogoll L, Azzarello-Burri S, Sheth F, Datar C, Verma IC, Puri RD, Zollino M, Bachmann-Gagescu R, Niedrist D, Papik M, Figueiro-Silva J, Masood R, Zweier M, Kraemer D, Lincoln S, Rodan L; Undiagnosed Diseases Network (UDN); Passemard S, Drunat S, Verloes A, Horn AHC, Sticht H, Steinfeld R, Plecko B, Latal B, Jenni O, Asadollahi R, Rauch A. Elucidation of the phenotypic spectrum and genetic landscape in primary and secondary microcephaly. Genet Med. 2019 Sep;21(9):2043-2058. doi: 10.1038/s41436-019-0464-7. Epub 2019 Mar 7. PMID 30842647
- [Background] Bainbridge MN, Mazumder A, Ogasawara D, Abou Jamra R, Bernard G, Bertini E, Burglen L, Cope H, Crawford A, Derksen A, Dure L, Gantz E, Koch-Hogrebe M, Hurst ACE, Mahida S, Marshall P, Micalizzi A, Novelli A, Peng H; Rady Children's Institute for Genomic Medicine; Rodriguez D, Robbins SL, Rutledge SL, Scalise R, Schliesske S, Shashi V, Srivastava S, Thiffault I, Topol S; Undiagnosed Disease Network; Qebibo L, Wieczorek D, Cravatt B, Haricharan S, Torkamani A, Friedman J. Endocannabinoid dysfunction in neurological disease: neuro-ocular DAGLA-related syndrome. Brain. 2022 Oct 21;145(10):3383-3390. doi: 10.1093/brain/awac223. PMID 35737950
- [Background] Zastrow DB, Zornio PA, Dries A, Kohler J, Fernandez L, Waggott D, Walkiewicz M, Eng CM, Manning MA, Farrelly E; Undiagnosed Diseases Network; Fisher PG, Ashley EA, Bernstein JA, Wheeler MT. Exome sequencing identifies de novo pathogenic variants in FBN1 and TRPS1 in a patient with a complex connective tissue phenotype. Cold Spring Harb Mol Case Stud. 2017 Jan;3(1):a001388. doi: 10.1101/mcs.a001388. PMID 28050602
- [Background] Sullivan JA, Schoch K, Spillmann RC, Shashi V. Exome/Genome Sequencing in Undiagnosed Syndromes. Annu Rev Med. 2023 Jan 27;74:489-502. doi: 10.1146/annurev-med-042921-110721. PMID 36706750
- [Background] Zou F, McWalter K, Schmidt L, Decker A, Picker JD, Lincoln S, Sweetser DA, Briere LC, Harini C; Members of the Undiagnosed Diseases Network; Marsh E, Medne L, Wang RY, Leydiker K, Mower A, Visser G, Cuppen I, van Gassen KL, van der Smagt J, Yousaf A, Tennison M, Shanmugham A, Butler E, Richard G, McKnight D. Expanding the phenotypic spectrum of GABRG2 variants: a recurrent GABRG2 missense variant associated with a severe phenotype. J Neurogenet. 2017 Mar-Jun;31(1-2):30-36. doi: 10.1080/01677063.2017.1315417. Epub 2017 May 2. PMID 28460589
- [Background] Machol K, Rousseau J, Ehresmann S, Garcia T, Nguyen TTM, Spillmann RC, Sullivan JA, Shashi V, Jiang YH, Stong N, Fiala E, Willing M, Pfundt R, Kleefstra T, Cho MT, McLaughlin H, Rosello Piera M, Orellana C, Martinez F, Caro-Llopis A, Monfort S, Roscioli T, Nixon CY, Buckley MF, Turner A, Jones WD, van Hasselt PM, Hofstede FC, van Gassen KLI, Brooks AS, van Slegtenhorst MA, Lachlan K, Sebastian J, Madan-Khetarpal S, Sonal D, Sakkubai N, Thevenon J, Faivre L, Maurel A, Petrovski S, Krantz ID, Tarpinian JM, Rosenfeld JA, Lee BH; Undiagnosed Diseases Network; Campeau PM. Expanding the Spectrum of BAF-Related Disorders: De Novo Variants in SMARCC2 Cause a Syndrome with Intellectual Disability and Developmental Delay. Am J Hum Genet. 2019 Jan 3;104(1):164-178. doi: 10.1016/j.ajhg.2018.11.007. Epub 2018 Dec 20. PMID 30580808
- [Background] Mis EK, Sega AG, Signer RH, Cartwright T, Ji W, Martinez-Agosto JA, Nelson SF, Palmer CGS, Lee H, Mitzelfelt T, Konstantino M; Undiagnosed Diseases Network; Jeffries L, Khokha MK, Marco E, Martin MG, Lakhani SA. Expansion of NEUROD2 phenotypes to include developmental delay without seizures. Am J Med Genet A. 2021 Apr;185(4):1076-1080. doi: 10.1002/ajmg.a.62064. Epub 2021 Jan 13. PMID 33438828
- [Background] Kumar A, Zastrow DB, Kravets EJ, Beleford D, Ruzhnikov MRZ, Grove ME, Dries AM, Kohler JN, Waggott DM, Yang Y, Huang Y; Undiagnosed Diseases Network; Mackenzie KM, Eng CM, Fisher PG, Ashley EA, Teng JM, Stevenson DA, Shieh JT, Wheeler MT, Bernstein JA. Extracutaneous manifestations in phacomatosis cesioflammea and cesiomarmorata: Case series and literature review. Am J Med Genet A. 2019 Jun;179(6):966-977. doi: 10.1002/ajmg.a.61134. Epub 2019 Mar 28. PMID 30920161
- [Background] Shibao CA, Joos K, Phillips JA 3rd, Cogan J, Newman JH, Hamid R, Meiler J, Capra J, Sheehan J, Vetrini F, Yang Y, Black B, Diedrich A, Roberston D, Biaggioni I. Familial Autonomic Ganglionopathy Caused by Rare CHRNA3 Genetic Variants. Neurology. 2021 Jul 13;97(2):e145-e155. doi: 10.1212/WNL.0000000000012143. Epub 2021 May 4. PMID 33947782
- [Background] Studwell CM, Glanton E; Undiagnosed Diseases Network; Sinsheimer JS, Palmer CGS, LeBlanc K. Family genetic result communication in rare and undiagnosed disease communities: Understanding the practice. J Genet Couns. 2021 Apr;30(2):439-447. doi: 10.1002/jgc4.1329. Epub 2020 Oct 27. PMID 33108040
- [Background] Yates J, Gutierrez-Sacristan A, Jouhet V, LeBlanc K, Esteves C; Undiagnosed Diseases Network; DeSain TN, Benik N, Stedman J, Palmer N, Mellon G, Kohane I, Avillach P. Finding commonalities in rare diseases through the undiagnosed diseases network. J Am Med Inform Assoc. 2021 Jul 30;28(8):1694-1702. doi: 10.1093/jamia/ocab050. PMID 34009343
- [Background] Stergachis AB, Blue EE, Gillentine MA, Wang LK, Schwarze U, Cortes AS, Ranchalis J, Allworth A, Bland AE, Chanprasert S, Chen J, Doherty D, Folta AB, Glass I, Horike-Pyne M, Huang AY, Khan AT, Leppig KA, Miller DE, Mirzaa G, Parhin A, Raskind W, Rosenthal EA, Sheppeard S, Strohbehn S, Sybert VP, Tran TT, Wener M; University of Washington Center for Mendelian Genomics (UW-CMG), Undiagnosed Diseases Network (UDN); Byers PH, Nelson SF, Bamshad MJ, Dipple KM, Jarvik GP, Hoppins S, Hisama FM. Full-length isoform sequencing for resolving the molecular basis of Charcot-Marie-Tooth 2A. bioRxiv [Preprint]. 2023 Feb 7:2023.02.07.526487. doi: 10.1101/2023.02.07.526487. PMID 36798371
- [Background] Boulin T, Itani O, El Mouridi S, Leclercq-Blondel A, Gendrel M, Macnamara E, Soldatos A, Murphy JL, Gorman MP, Lindsey A, Shimada S, Turner D, Silverman GA, Baldridge D; Undiagnosed Diseases Network; Malicdan MC, Schedl T, Pak SC. Functional analysis of a de novo variant in the neurodevelopment and generalized epilepsy disease gene NBEA. Mol Genet Metab. 2021 Sep-Oct;134(1-2):195-202. doi: 10.1016/j.ymgme.2021.07.013. Epub 2021 Aug 9. PMID 34412939
- [Background] Fielder SM, Rosenfeld JA, Burrage LC, Emrick L, Lalani S, Attali R, Bembenek JN, Hoang H, Baldridge D, Silverman GA; Undiagnosed Diseases Network; Schedl T, Pak SC. Functional analysis of a novel de novo variant in PPP5C associated with microcephaly, seizures, and developmental delay. Mol Genet Metab. 2022 May;136(1):65-73. doi: 10.1016/j.ymgme.2022.03.007. Epub 2022 Mar 22. PMID 35361529
- [Background] Liu N, Schoch K, Luo X, Pena LDM, Bhavana VH, Kukolich MK, Stringer S, Powis Z, Radtke K, Mroske C, Deak KL, McDonald MT, McConkie-Rosell A, Markert ML, Kranz PG, Stong N, Need AC, Bick D, Amaral MD, Worthey EA, Levy S; Undiagnosed Diseases Network (UDN); Wangler MF, Bellen HJ, Shashi V, Yamamoto S. Functional variants in TBX2 are associated with a syndromic cardiovascular and skeletal developmental disorder. Hum Mol Genet. 2018 Jul 15;27(14):2454-2465. doi: 10.1093/hmg/ddy146. PMID 29726930
- [Background] Tan QK, Cope H, Spillmann RC, Stong N, Jiang YH, McDonald MT, Rothman JA, Butler MW, Frush DP, Lachman RS, Lee B, Bacino CA, Bonner MJ, McCall CM, Pendse AA, Walley N; Undiagnosed Diseases Network; Shashi V, Pena LDM. Further evidence for the involvement of EFL1 in a Shwachman-Diamond-like syndrome and expansion of the phenotypic features. Cold Spring Harb Mol Case Stud. 2018 Oct 1;4(5):a003046. doi: 10.1101/mcs.a003046. Print 2018 Oct. PMID 29970384
- [Background] Kozycki CT, Kodati S, Huryn L, Wang H, Warner BM, Jani P, Hammoud D, Abu-Asab MS, Jittayasothorn Y, Mattapallil MJ, Tsai WL, Ullah E, Zhou P, Tian X, Soldatos A, Moutsopoulos N, Kao-Hsieh M, Heller T, Cowen EW, Lee CR, Toro C, Kalsi S, Khavandgar Z, Baer A, Beach M, Long Priel D, Nehrebecky M, Rosenzweig S, Romeo T, Deuitch N, Brenchley L, Pelayo E, Zein W, Sen N, Yang AH, Farley G, Sweetser DA, Briere L, Yang J, de Oliveira Poswar F, Schwartz IVD, Silva Alves T, Dusser P, Kone-Paut I, Touitou I, Titah SM, van Hagen PM, van Wijck RTA, van der Spek PJ, Yano H, Benneche A, Apalset EM, Jansson RW, Caspi RR, Kuhns DB, Gadina M, Takada H, Ida H, Nishikomori R, Verrecchia E, Sangiorgi E, Manna R, Brooks BP, Sobrin L, Hufnagel RB, Beck D, Shao F, Ombrello AK, Aksentijevich I, Kastner DL; Undiagnosed Diseases Network. Gain-of-function mutations in ALPK1 cause an NF-kappaB-mediated autoinflammatory disease: functional assessment, clinical phenotyping and disease course of patients with ROSAH syndrome. Ann Rheum Dis. 2022 Oct;81(10):1453-1464. doi: 10.1136/annrheumdis-2022-222629. Epub 2022 Jul 22. PMID 35868845
- [Background] Sharma R, Sahoo SS, Honda M, Granger SL, Goodings C, Sanchez L, Kunstner A, Busch H, Beier F, Pruett-Miller SM, Valentine MB, Fernandez AG, Chang TC, Geli V, Churikov D, Hirschi S, Pastor VB, Boerries M, Lauten M, Kelaidi C, Cooper MA, Nicholas S, Rosenfeld JA, Polychronopoulou S, Kannengiesser C, Saintome C, Niemeyer CM, Revy P, Wold MS, Spies M, Erlacher M, Coulon S, Wlodarski MW. Gain-of-function mutations in RPA1 cause a syndrome with short telomeres and somatic genetic rescue. Blood. 2022 Feb 17;139(7):1039-1051. doi: 10.1182/blood.2021011980. PMID 34767620
- [Background] Shieh C, Jones N, Vanle B, Au M, Huang AY, Silva APG, Lee H, Douine ED, Otero MG, Choi A, Grand K, Taff IP, Delgado MR, Hajianpour MJ, Seeley A, Rohena L, Vernon H, Gripp KW, Vergano SA, Mahida S, Naidu S, Sousa AB, Wain KE, Challman TD, Beek G, Basel D, Ranells J, Smith R, Yusupov R, Freckmann ML, Ohden L, Davis-Keppen L, Chitayat D, Dowling JJ, Finkel R, Dauber A, Spillmann R, Pena LDM; Undiagnosed Diseases Network; Metcalfe K, Splitt M, Lachlan K, McKee SA, Hurst J, Fitzpatrick DR, Morton JEV, Cox H, Venkateswaran S, Young JI, Marsh ED, Nelson SF, Martinez JA, Graham JM Jr, Kini U, Mackay JP, Pierson TM. GATAD2B-associated neurodevelopmental disorder (GAND): clinical and molecular insights into a NuRD-related disorder. Genet Med. 2020 May;22(5):878-888. doi: 10.1038/s41436-019-0747-z. Epub 2020 Jan 17. PMID 31949314
- [Background] Scala M, Bradley CA, Howe JL, Trost B, Salazar NB, Shum C, Reuter MS, MacDonald JR, Ko SY, Frankland PW, Granger L, Anadiotis G, Pullano V, Brusco A, Keller R, Parisotto S, Pedro HF, Lusk L, McDonnell PP, Helbig I, Mullegama SV; Undiagnosed Diseases Network; Douine ED, Russell BE, Nelson SF, Zara F, Scherer SW. Genetic variants in DDX53 contribute to Autism Spectrum Disorder associated with the Xp22.11 locus. medRxiv [Preprint]. 2023 Dec 27:2023.12.21.23300383. doi: 10.1101/2023.12.21.23300383. PMID 38234782
- [Background] Borja N, Bivona S, Peart LS, Johnson B, Gonzalez J, Barbouth D, Moore H, Guo S; Undiagnosed Disease Network; Bademci G, Tekin M. Genome sequencing reveals novel noncoding variants in PLA2G6 and LMNB1 causing progressive neurologic disease. Mol Genet Genomic Med. 2022 Apr;10(4):e1892. doi: 10.1002/mgg3.1892. Epub 2022 Mar 5. PMID 35247231
- [Background] Halley MC, Young JL, Tang C, Mintz KT, Lucas-Griffin S, Maghiro A, Ashley EA, Tabor HK; Undiagnosed Diseases Network. Genomics Research with Undiagnosed Children: Ethical Challenges at the Boundaries of Research and Clinical Care. J Pediatr. 2023 Oct;261:113537. doi: 10.1016/j.jpeds.2023.113537. Epub 2023 Jun 2. PMID 37271495
- [Background] Jordan VK, Fregeau B, Ge X, Giordano J, Wapner RJ, Balci TB, Carter MT, Bernat JA, Moccia AN, Srivastava A, Martin DM, Bielas SL, Pappas J, Svoboda MD, Rio M, Boddaert N, Cantagrel V, Lewis AM, Scaglia F; Undiagnosed Diseases Network; Kohler JN, Bernstein JA, Dries AM, Rosenfeld JA, DeFilippo C, Thorson W, Yang Y, Sherr EH, Bi W, Scott DA. Genotype-phenotype correlations in individuals with pathogenic RERE variants. Hum Mutat. 2018 May;39(5):666-675. doi: 10.1002/humu.23400. Epub 2018 Jan 25. PMID 29330883
- [Background] Borja N, Borjas-Mendoza P, Bivona S, Peart L, Gonzalez J, Johnson BK, Guo S, Yusupov R; Undiagnosed Diseases Network; Bademci G, Tekin M. H4C5 missense variant leads to a neurodevelopmental phenotype overlapping with Angelman syndrome. Am J Med Genet A. 2023 Jul;191(7):1911-1916. doi: 10.1002/ajmg.a.63193. Epub 2023 Mar 29. PMID 36987712
- [Background] Bosticardo M, Yamazaki Y, Cowan J, Giardino G, Corsino C, Scalia G, Prencipe R, Ruffner M, Hill DA, Sakovich I, Yemialyanava I, Tam JS, Padem N, Elder ME, Sleasman JW, Perez E, Niebur H, Seroogy CM, Sharapova S, Gebbia J, Kleiner GI, Peake J, Abbott JK, Gelfand EW, Crestani E, Biggs C, Butte MJ, Hartog N, Hayward A, Chen K, Heimall J, Seeborg F, Bartnikas LM, Cooper MA, Pignata C, Bhandoola A, Notarangelo LD. Heterozygous FOXN1 Variants Cause Low TRECs and Severe T Cell Lymphopenia, Revealing a Crucial Role of FOXN1 in Supporting Early Thymopoiesis. Am J Hum Genet. 2019 Sep 5;105(3):549-561. doi: 10.1016/j.ajhg.2019.07.014. Epub 2019 Aug 22. PMID 31447097
- [Background] Ravenscroft TA, Phillips JB, Fieg E, Bajikar SS, Peirce J, Wegner J, Luna AA, Fox EJ, Yan YL, Rosenfeld JA, Zirin J, Kanca O; Undiagnosed Diseases Network; Benke PJ, Cameron ES, Strehlow V, Platzer K, Jamra RA, Klockner C, Osmond M, Licata T, Rojas S, Dyment D, Chong JSC, Lincoln S, Stoler JM, Postlethwait JH, Wangler MF, Yamamoto S, Krier J, Westerfield M, Bellen HJ. Heterozygous loss-of-function variants significantly expand the phenotypes associated with loss of GDF11. Genet Med. 2021 Oct;23(10):1889-1900. doi: 10.1038/s41436-021-01216-8. Epub 2021 Jun 10. PMID 34113007
- [Background] Ganapathi M, Matsuoka LS, March M, Li D, Brokamp E, Benito-Sanz S, White SM, Lachlan K, Ahimaz P, Sewda A, Bastarache L, Thomas-Wilson A, Stoler JM, Bramswig NC, Baptista J, Stals K, Demurger F, Cogne B, Isidor B, Bedeschi MF, Peron A, Amiel J, Zackai E, Schacht JP, Iglesias AD, Morton J, Schmetz A; Undiagnosed Diseases Network; Seidel V, Lucia S, Baskin SM, Thiffault I, Cogan JD, Gordon CT, Chung WK, Bowdin S, Bhoj E. Heterozygous rare variants in NR2F2 cause a recognizable multiple congenital anomaly syndrome with developmental delays. Eur J Hum Genet. 2023 Oct;31(10):1117-1124. doi: 10.1038/s41431-023-01434-5. Epub 2023 Jul 27. PMID 37500725
- [Background] Poli MC, Ebstein F, Nicholas SK, de Guzman MM, Forbes LR, Chinn IK, Mace EM, Vogel TP, Carisey AF, Benavides F, Coban-Akdemir ZH, Gibbs RA, Jhangiani SN, Muzny DM, Carvalho CMB, Schady DA, Jain M, Rosenfeld JA, Emrick L, Lewis RA, Lee B; Undiagnosed Diseases Network members; Zieba BA, Kury S, Kruger E, Lupski JR, Bostwick BL, Orange JS. Heterozygous Truncating Variants in POMP Escape Nonsense-Mediated Decay and Cause a Unique Immune Dysregulatory Syndrome. Am J Hum Genet. 2018 Jun 7;102(6):1126-1142. doi: 10.1016/j.ajhg.2018.04.010. Epub 2018 May 24. PMID 29805043
- [Background] Shashi V, Geist J, Lee Y, Yoo Y, Shin U, Schoch K, Sullivan J, Stong N, Smith E, Jasien J, Kranz P; Undiagnosed Diseases Network; Lee Y, Shin YB, Wright NT, Choi M, Kontrogianni-Konstantopoulos A. Heterozygous variants in MYBPC1 are associated with an expanded neuromuscular phenotype beyond arthrogryposis. Hum Mutat. 2019 Aug;40(8):1115-1126. doi: 10.1002/humu.23760. Epub 2019 May 5. PMID 31264822
- [Background] Mueller AA, Sasaki T, Keegan JW, Nguyen JP, Griffith A, Horisberger AM, Licata T, Fieg E, Cao Y, Elahee M, Marks KE, Simmons DP, Briere LC, Cobban LA, Pallais JC, High FA, Walker MA, Linnoila JJ, Sparks JA, Holers VM, Costenbader KH; Undiagnosed Diseases Network; Sweetser DA, Krier JB, Loscalzo J, Lederer JA, Rao DA. High-dimensional immunophenotyping reveals immune cell aberrations in patients with undiagnosed inflammatory and autoimmune diseases. J Clin Invest. 2023 Dec 15;133(24):e169619. doi: 10.1172/JCI169619. No abstract available. PMID 37874643
- [Background] Bryant L, Li D, Cox SG, Marchione D, Joiner EF, Wilson K, Janssen K, Lee P, March ME, Nair D, Sherr E, Fregeau B, Wierenga KJ, Wadley A, Mancini GMS, Powell-Hamilton N, van de Kamp J, Grebe T, Dean J, Ross A, Crawford HP, Powis Z, Cho MT, Willing MC, Manwaring L, Schot R, Nava C, Afenjar A, Lessel D, Wagner M, Klopstock T, Winkelmann J, Catarino CB, Retterer K, Schuette JL, Innis JW, Pizzino A, Luttgen S, Denecke J, Strom TM, Monaghan KG; DDD Study; Yuan ZF, Dubbs H, Bend R, Lee JA, Lyons MJ, Hoefele J, Gunthner R, Reutter H, Keren B, Radtke K, Sherbini O, Mrokse C, Helbig KL, Odent S, Cogne B, Mercier S, Bezieau S, Besnard T, Kury S, Redon R, Reinson K, Wojcik MH, Ounap K, Ilves P, Innes AM, Kernohan KD; Care4Rare Canada Consortium; Costain G, Meyn MS, Chitayat D, Zackai E, Lehman A, Kitson H; CAUSES Study; Martin MG, Martinez-Agosto JA; Undiagnosed Diseases Network; Nelson SF, Palmer CGS, Papp JC, Parker NH, Sinsheimer JS, Vilain E, Wan J, Yoon AJ, Zheng A, Brimble E, Ferrero GB, Radio FC, Carli D, Barresi S, Brusco A, Tartaglia M, Thomas JM, Umana L, Weiss MM, Gotway G, Stuurman KE, Thompson ML, McWalter K, Stumpel CTRM, Stevens SJC, Stegmann APA, Tveten K, Vollo A, Prescott T, Fagerberg C, Laulund LW, Larsen MJ, Byler M, Lebel RR, Hurst AC, Dean J, Schrier Vergano SA, Norman J, Mercimek-Andrews S, Neira J, Van Allen MI, Longo N, Sellars E, Louie RJ, Cathey SS, Brokamp E, Heron D, Snyder M, Vanderver A, Simon C, de la Cruz X, Padilla N, Crump JG, Chung W, Garcia B, Hakonarson HH, Bhoj EJ. Histone H3.3 beyond cancer: Germline mutations in Histone 3 Family 3A and 3B cause a previously unidentified neurodegenerative disorder in 46 patients. Sci Adv. 2020 Dec 2;6(49):eabc9207. doi: 10.1126/sciadv.abc9207. Print 2020 Dec. PMID 33268356
- [Background] Niggl E, Bouman A, Briere LC, Hoogenboezem RM, Wallaard I, Park J, Admard J, Wilke M, Harris-Mostert EDRO, Elgersma M, Bain J, Balasubramanian M, Banka S, Benke PJ, Bertrand M, Blesson AE, Clayton-Smith J, Ellingford JM, Gillentine MA, Goodloe DH, Haack TB, Jain M, Krantz I, Luu SM, McPheron M, Muss CL, Raible SE, Robin NH, Spiller M, Starling S, Sweetser DA, Thiffault I, Vetrini F, Witt D, Woods E, Zhou D; Genomics England Research Consortium; Undiagnosed Diseases Network; Elgersma Y, van Esbroeck ACM. HNRNPC haploinsufficiency affects alternative splicing of intellectual disability-associated genes and causes a neurodevelopmental disorder. Am J Hum Genet. 2023 Aug 3;110(8):1414-1435. doi: 10.1016/j.ajhg.2023.07.005. PMID 37541189
- [Background] Davids M, Menezes M, Guo Y, McLean SD, Hakonarson H, Collins F, Worgan L, Billington CJ Jr, Maric I, Littlejohn RO, Onyekweli T, Members Of The Udn, Adams DR, Tifft CJ, Gahl WA, Wolfe LA, Christodoulou J, Malicdan MCV. Homozygous splice-variants in human ARV1 cause GPI-anchor synthesis deficiency. Mol Genet Metab. 2020 May;130(1):49-57. doi: 10.1016/j.ymgme.2020.02.005. Epub 2020 Feb 10. PMID 32165008
- [Background] Bonder MJ, Smail C, Gloudemans MJ, Fresard L, Jakubosky D, D'Antonio M, Li X, Ferraro NM, Carcamo-Orive I, Mirauta B, Seaton DD, Cai N, Vakili D, Horta D, Zhao C, Zastrow DB, Bonner DE; HipSci Consortium; iPSCORE consortium; Undiagnosed Diseases Network; PhLiPS consortium; Wheeler MT, Kilpinen H, Knowles JW, Smith EN, Frazer KA, Montgomery SB, Stegle O. Identification of rare and common regulatory variants in pluripotent cells using population-scale transcriptomics. Nat Genet. 2021 Mar;53(3):313-321. doi: 10.1038/s41588-021-00800-7. Epub 2021 Mar 4. PMID 33664507
- [Background] Fresard L, Smail C, Ferraro NM, Teran NA, Li X, Smith KS, Bonner D, Kernohan KD, Marwaha S, Zappala Z, Balliu B, Davis JR, Liu B, Prybol CJ, Kohler JN, Zastrow DB, Reuter CM, Fisk DG, Grove ME, Davidson JM, Hartley T, Joshi R, Strober BJ, Utiramerur S; Undiagnosed Diseases Network; Care4Rare Canada Consortium; Lind L, Ingelsson E, Battle A, Bejerano G, Bernstein JA, Ashley EA, Boycott KM, Merker JD, Wheeler MT, Montgomery SB. Identification of rare-disease genes using blood transcriptome sequencing and large control cohorts. Nat Med. 2019 Jun;25(6):911-919. doi: 10.1038/s41591-019-0457-8. Epub 2019 Jun 3. PMID 31160820
- [Background] Mukherjee S, Cogan JD, Newman JH, Phillips JA 3rd, Hamid R; Undiagnosed Diseases Network; Meiler J, Capra JA. Identifying digenic disease genes via machine learning in the Undiagnosed Diseases Network. Am J Hum Genet. 2021 Oct 7;108(10):1946-1963. doi: 10.1016/j.ajhg.2021.08.010. Epub 2021 Sep 15. PMID 34529933
- [Background] Newman JH, Shaver A, Sheehan JH, Mallal S, Stone JH, Pillai S, Bastarache L, Riebau D, Allard-Chamard H, Stone WM, Perugino C, Pilkinton M, Smith SA, McDonnell WJ, Capra JA, Meiler J, Cogan J, Xing K, Mahajan VS, Mattoo H, Hamid R, Phillips JA 3rd; Undiagnosed Disease Network. IgG4-related disease: Association with a rare gene variant expressed in cytotoxic T cells. Mol Genet Genomic Med. 2019 Jun;7(6):e686. doi: 10.1002/mgg3.686. Epub 2019 Apr 16. PMID 30993913
- [Background] Ungar RA, Goddard PC, Jensen TD, Degalez F, Smith KS, Jin CA; Undiagnosed Diseases Network; Bonner DE, Bernstein JA, Wheeler MT, Montgomery SB. Impact of genome build on RNA-seq interpretation and diagnostics. medRxiv [Preprint]. 2024 Jan 12:2024.01.11.24301165. doi: 10.1101/2024.01.11.24301165. PMID 38260490
- [Background] Splinter K, Hull SC, Holm IA, McDonough TL, Wise AL, Ramoni RB; Members of the Undiagnosed Diseases Network. Implementing the Single Institutional Review Board Model: Lessons from the Undiagnosed Diseases Network. Clin Transl Sci. 2018 Jan;11(1):28-31. doi: 10.1111/cts.12512. Epub 2017 Oct 23. No abstract available. PMID 28945957
- [Background] Harnish JM, Deal SL, Chao HT, Wangler MF, Yamamoto S. In Vivo Functional Study of Disease-associated Rare Human Variants Using Drosophila. J Vis Exp. 2019 Aug 20;(150):10.3791/59658. doi: 10.3791/59658. PMID 31498321
- [Background] Marcogliese PC, Shashi V, Spillmann RC, Stong N, Rosenfeld JA, Koenig MK, Martinez-Agosto JA, Herzog M, Chen AH, Dickson PI, Lin HJ, Vera MU, Salamon N, Graham JM Jr, Ortiz D, Infante E, Steyaert W, Dermaut B, Poppe B, Chung HL, Zuo Z, Lee PT, Kanca O, Xia F, Yang Y, Smith EC, Jasien J, Kansagra S, Spiridigliozzi G, El-Dairi M, Lark R, Riley K, Koeberl DD, Golden-Grant K; Program for Undiagnosed Diseases (UD-PrOZA); Undiagnosed Diseases Network; Yamamoto S, Wangler MF, Mirzaa G, Hemelsoet D, Lee B, Nelson SF, Goldstein DB, Bellen HJ, Pena LDM. IRF2BPL Is Associated with Neurological Phenotypes. Am J Hum Genet. 2018 Aug 2;103(2):245-260. doi: 10.1016/j.ajhg.2018.07.006. Epub 2018 Jul 26. PMID 30057031
- [Background] Kilich G, Hassey K, Behrens EM, Falk M, Vanderver A, Rader DJ, Cahill PJ, Raper A, Zhang Z, Westerfer D, Jadhav T, Conlin L, Izumi K, Rajagopalan R, Sullivan KE; UDN Consortium. Kagami Ogata syndrome: a small deletion refines critical region for imprinting. NPJ Genom Med. 2024 Jan 11;9(1):5. doi: 10.1038/s41525-023-00389-2. PMID 38212313
- [Background] Macnamara EF, Koehler AE, D'Souza P, Estwick T, Lee P, Vezina G; Undiagnosed Diseases Network; Fauni H, Braddock SR, Torti E, Holt JM, Sharma P, Malicdan MCV, Tifft CJ. Kilquist syndrome: A novel syndromic hearing loss disorder caused by homozygous deletion of SLC12A2. Hum Mutat. 2019 May;40(5):532-538. doi: 10.1002/humu.23722. Epub 2019 Mar 12. PMID 30740830
- [Background] Cif L, Demailly D, Lin JP, Barwick KE, Sa M, Abela L, Malhotra S, Chong WK, Steel D, Sanchis-Juan A, Ngoh A, Trump N, Meyer E, Vasques X, Rankin J, Allain MW, Applegate CD, Attaripour Isfahani S, Baleine J, Balint B, Bassetti JA, Baple EL, Bhatia KP, Blanchet C, Burglen L, Cambonie G, Seng EC, Bastaraud SC, Cyprien F, Coubes C, d'Hardemare V; Deciphering Developmental Disorders Study; Doja A, Dorison N, Doummar D, Dy-Hollins ME, Farrelly E, Fitzpatrick DR, Fearon C, Fieg EL, Fogel BL, Forman EB, Fox RG; Genomics England Research Consortium; Gahl WA, Galosi S, Gonzalez V, Graves TD, Gregory A, Hallett M, Hasegawa H, Hayflick SJ, Hamosh A, Hully M, Jansen S, Jeong SY, Krier JB, Krystal S, Kumar KR, Laurencin C, Lee H, Lesca G, Francois LL, Lynch T, Mahant N, Martinez-Agosto JA, Milesi C, Mills KA, Mondain M, Morales-Briceno H; NIHR BioResource; Ostergaard JR, Pal S, Pallais JC, Pavillard F, Perrigault PF, Petersen AK, Polo G, Poulen G, Rinne T, Roujeau T, Rogers C, Roubertie A, Sahagian M, Schaefer E, Selim L, Selway R, Sharma N, Signer R, Soldatos AG, Stevenson DA, Stewart F, Tchan M; Undiagnosed Diseases Network; Verma IC, de Vries BBA, Wilson JL, Wong DA, Zaitoun R, Zhen D, Znaczko A, Dale RC, de Gusmao CM, Friedman J, Fung VSC, King MD, Mohammad SS, Rohena L, Waugh JL, Toro C, Raymond FL, Topf M, Coubes P, Gorman KM, Kurian MA. KMT2B-related disorders: expansion of the phenotypic spectrum and long-term efficacy of deep brain stimulation. Brain. 2020 Dec 5;143(11):3242-3261. doi: 10.1093/brain/awaa304. PMID 33150406
- [Background] Burdick KJ, Cogan JD, Rives LC, Robertson AK, Koziura ME, Brokamp E, Duncan L, Hannig V, Pfotenhauer J, Vanzo R, Paul MS, Bican A, Morgan T, Duis J, Newman JH, Hamid R, Phillips JA 3rd; Undiagnosed Diseases Network. Limitations of exome sequencing in detecting rare and undiagnosed diseases. Am J Med Genet A. 2020 Jun;182(6):1400-1406. doi: 10.1002/ajmg.a.61558. Epub 2020 Mar 19. PMID 32190976
- [Background] Beck DB, Basar MA, Asmar AJ, Thompson JJ, Oda H, Uehara DT, Saida K, Pajusalu S, Talvik I, D'Souza P, Bodurtha J, Mu W, Baranano KW, Miyake N, Wang R, Kempers M, Tamada T, Nishimura Y, Okada S, Kosho T, Dale R, Mitra A, Macnamara E; Undiagnosed Diseases Network; Matsumoto N, Inazawa J, Walkiewicz M, Ounap K, Tifft CJ, Aksentijevich I, Kastner DL, Rocha PP, Werner A. Linkage-specific deubiquitylation by OTUD5 defines an embryonic pathway intolerant to genomic variation. Sci Adv. 2021 Jan 20;7(4):eabe2116. doi: 10.1126/sciadv.abe2116. Print 2021 Jan. PMID 33523931
- [Background] Pena LDM, Jiang YH, Schoch K, Spillmann RC, Walley N, Stong N, Rapisardo Horn S, Sullivan JA, McConkie-Rosell A, Kansagra S, Smith EC, El-Dairi M, Bellet J, Keels MA, Jasien J, Kranz PG, Noel R, Nagaraj SK, Lark RK, Wechsler DSG, Del Gaudio D, Leung ML, Hendon LG, Parker CC, Jones KL; Undiagnosed Diseases Network Members; Goldstein DB, Shashi V. Looking beyond the exome: a phenotype-first approach to molecular diagnostic resolution in rare and undiagnosed diseases. Genet Med. 2018 Apr;20(4):464-469. doi: 10.1038/gim.2017.128. Epub 2017 Sep 14. PMID 28914269
- [Background] Marcogliese PC, Dutta D, Ray SS, Dang NDP, Zuo Z, Wang Y, Lu D, Fazal F, Ravenscroft TA, Chung H, Kanca O, Wan J, Douine ED, Network UD, Pena LDM, Yamamoto S, Nelson SF, Might M, Meyer KC, Yeo NC, Bellen HJ. Loss of IRF2BPL impairs neuronal maintenance through excess Wnt signaling. Sci Adv. 2022 Jan 21;8(3):eabl5613. doi: 10.1126/sciadv.abl5613. Epub 2022 Jan 19. PMID 35044823
- [Background] Accogli A, Lu S, Musante I, Scudieri P, Rosenfeld JA, Severino M, Baldassari S, Iacomino M, Riva A, Balagura G, Piccolo G, Minetti C, Roberto D, Xia F, Razak R, Lawrence E, Hussein M, Chang EY, Holick M, Cali E, Aliberto E, De-Sarro R, Gambardella A, Network UD, Group SS, Emrick L, McCaffery PJA, Clagett-Dame M, Marcogliese PC, Bellen HJ, Lalani SR, Zara F, Striano P, Salpietro V. Loss of Neuron Navigator 2 Impairs Brain and Cerebellar Development. Cerebellum. 2023 Apr;22(2):206-222. doi: 10.1007/s12311-022-01379-3. Epub 2022 Feb 26. PMID 35218524
- [Background] Shashi V, Magiera MM, Klein D, Zaki M, Schoch K, Rudnik-Schoneborn S, Norman A, Lopes Abath Neto O, Dusl M, Yuan X, Bartesaghi L, De Marco P, Alfares AA, Marom R, Arold ST, Guzman-Vega FJ, Pena LD, Smith EC, Steinlin M, Babiker MO, Mohassel P, Foley AR, Donkervoort S, Kaur R, Ghosh PS, Stanley V, Musaev D, Nava C, Mignot C, Keren B, Scala M, Tassano E, Picco P, Doneda P, Fiorillo C, Issa MY, Alassiri A, Alahmad A, Gerard A, Liu P, Yang Y, Ertl-Wagner B, Kranz PG, Wentzensen IM, Stucka R, Stong N, Allen AS, Goldstein DB; Undiagnosed Diseases Network; Schoser B, Rosler KM, Alfadhel M, Capra V, Chrast R, Strom TM, Kamsteeg EJ, Bonnemann CG, Gleeson JG, Martini R, Janke C, Senderek J. Loss of tubulin deglutamylase CCP1 causes infantile-onset neurodegeneration. EMBO J. 2018 Dec 3;37(23):e100540. doi: 10.15252/embj.2018100540. Epub 2018 Nov 12. PMID 30420557
- [Background] Chung HL, Wangler MF, Marcogliese PC, Jo J, Ravenscroft TA, Zuo Z, Duraine L, Sadeghzadeh S, Li-Kroeger D, Schmidt RE, Pestronk A, Rosenfeld JA, Burrage L, Herndon MJ, Chen S; Members of Undiagnosed Diseases Network; Shillington A, Vawter-Lee M, Hopkin R, Rodriguez-Smith J, Henrickson M, Lee B, Moser AB, Jones RO, Watkins P, Yoo T, Mar S, Choi M, Bucelli RC, Yamamoto S, Lee HK, Prada CE, Chae JH, Vogel TP, Bellen HJ. Loss- or Gain-of-Function Mutations in ACOX1 Cause Axonal Loss via Different Mechanisms. Neuron. 2020 May 20;106(4):589-606.e6. doi: 10.1016/j.neuron.2020.02.021. Epub 2020 Mar 12. PMID 32169171
- [Background] AlAbdi L, Desbois M, Rusnac DV, Sulaiman RA, Rosenfeld JA, Lalani S, Murdock DR, Burrage LC; Undiagnosed Diseases Network; Billie Au PY, Towner S, Wilson WG, Wong L, Brunet T, Strobl-Wildemann G, Burton JE, Hoganson G, McWalter K, Begtrup A, Zarate YA, Christensen EL, Opperman KJ, Giles AC, Helaby R, Kania A, Zheng N, Grill B, Alkuraya FS. Loss-of-function variants in MYCBP2 cause neurobehavioural phenotypes and corpus callosum defects. Brain. 2023 Apr 19;146(4):1373-1387. doi: 10.1093/brain/awac364. PMID 36200388
- [Background] Lu J, Toro C, Adams DR; Undiagnosed Diseases Network; Moreno CAM, Lee WP, Leung YY, Harms MB, Vardarajan B, Heinzen EL. LUSTR: a new customizable tool for calling genome-wide germline and somatic short tandem repeat variants. BMC Genomics. 2024 Jan 26;25(1):115. doi: 10.1186/s12864-023-09935-9. PMID 38279154
- [Background] Nicoli ER, Weston MR, Hackbarth M, Becerril A, Larson A, Zein WM, Baker PR 2nd, Burke JD, Dorward H, Davids M, Huang Y, Adams DR, Zerfas PM, Chen D, Markello TC, Toro C, Wood T, Elliott G, Vu M; Undiagnosed Diseases Network; Zheng W, Garrett LJ, Tifft CJ, Gahl WA, Day-Salvatore DL, Mindell JA, Malicdan MCV. Lysosomal Storage and Albinism Due to Effects of a De Novo CLCN7 Variant on Lysosomal Acidification. Am J Hum Genet. 2019 Jun 6;104(6):1127-1138. doi: 10.1016/j.ajhg.2019.04.008. Epub 2019 May 30. PMID 31155284
- [Background] Amiri H, Kohane IS; Undiagnosed Diseases Network. Machine Learning of Patient Characteristics to Predict Admission Outcomes in the Undiagnosed Diseases Network. JAMA Netw Open. 2021 Feb 1;4(2):e2036220. doi: 10.1001/jamanetworkopen.2020.36220. PMID 33630084
- [Background] Koop K, Yuan W, Tessadori F, Rodriguez-Polanco WR, Grubbs J, Zhang B, Osmond M, Graham G, Sawyer S, Conboy E, Vetrini F, Treat K, Ploski R, Pienkowski VM, Klosowska A, Fieg E, Krier J, Mallebranche C, Alban Z, Aldinger KA, Ritter D, Macnamara E, Sullivan B, Herriges J, Alaimo JT, Helbig C, Ellis CA, van Eyk C, Gecz J, Farrugia D, Osei-Owusu I, Ades L, van den Boogaard MJ, Fuchs S, Bakker J, Duran K, Dawson ZD, Lindsey A, Huang H, Baldridge D, Silverman GA, Grant BD, Raizen D; Undiagnosed Diseases Network; van Haaften G, Pak SC, Rehmann H, Schedl T, van Hasselt P. Macrocephaly and developmental delay caused by missense variants in RAB5C. Hum Mol Genet. 2023 Oct 17;32(21):3063-3077. doi: 10.1093/hmg/ddad130. PMID 37552066
- [Background] Bhatia A, Mobley BC, Cogan J, Koziura ME, Brokamp E, Phillips J, Newman J; Undiagnosed Diseases Network (UDN); Moore SA, Hamid R; Members of the Undiagnosed Diseases Network. Magnetic Resonance Imaging characteristics in case of TOR1AIP1 muscular dystrophy. Clin Imaging. 2019 Nov-Dec;58:108-113. doi: 10.1016/j.clinimag.2019.06.010. Epub 2019 Jun 21. PMID 31299614
- [Background] Wang J, Al-Ouran R, Hu Y, Kim SY, Wan YW, Wangler MF, Yamamoto S, Chao HT, Comjean A, Mohr SE; UDN; Perrimon N, Liu Z, Bellen HJ. MARRVEL: Integration of Human and Model Organism Genetic Resources to Facilitate Functional Annotation of the Human Genome. Am J Hum Genet. 2017 Jun 1;100(6):843-853. doi: 10.1016/j.ajhg.2017.04.010. Epub 2017 May 11. PMID 28502612
- [Background] Emrick LT, Rosenfeld JA, Lalani SR, Jain M, Desai NK, Larson A, Kripps K, Vanderver A, Taft RJ, Bluske K, Perry D, Nagakura H, Immken LL, Burrage LC, Bacino CA, Belmont JW, Network UD, Lee B. Microdeletions excluding YWHAE and PAFAH1B1 cause a unique leukoencephalopathy: further delineation of the 17p13.3 microdeletion spectrum. Genet Med. 2019 Jul;21(7):1652-1656. doi: 10.1038/s41436-018-0358-0. Epub 2018 Dec 20. PMID 30568308
- [Background] Cope H, Spillmann R, Rosenfeld JA, Brokamp E, Signer R, Schoch K, Glanton E, Sullivan JA, Macnamara E, Lincoln S, Golden-Grant K; Undiagnosed Diseases Network; Orengo JP, Clark G, Burrage LC, Posey JE, Punetha J, Robertson A, Cogan J, Phillips JA 3rd, Martinez-Agosto J, Shashi V. Missed diagnoses: Clinically relevant lessons learned through medical mysteries solved by the Undiagnosed Diseases Network. Mol Genet Genomic Med. 2020 Oct;8(10):e1397. doi: 10.1002/mgg3.1397. Epub 2020 Jul 30. PMID 32730690
- [Background] Parenti I, Lehalle D, Nava C, Torti E, Leitao E, Person R, Mizuguchi T, Matsumoto N, Kato M, Nakamura K, de Man SA, Cope H, Shashi V; Undiagnosed Diseases Network; Friedman J, Joset P, Steindl K, Rauch A, Muffels I, van Hasselt PM, Petit F, Smol T, Le Guyader G, Bilan F, Sorlin A, Vitobello A, Philippe C, van de Laar IMBH, van Slegtenhorst MA, Campeau PM, Au PYB, Nakashima M, Saitsu H, Yamamoto T, Nomura Y, Louie RJ, Lyons MJ, Dobson A, Plomp AS, Motazacker MM, Kaiser FJ, Timberlake AT, Fuchs SA, Depienne C, Mignot C. Missense and truncating variants in CHD5 in a dominant neurodevelopmental disorder with intellectual disability, behavioral disturbances, and epilepsy. Hum Genet. 2021 Jul;140(7):1109-1120. doi: 10.1007/s00439-021-02283-2. Epub 2021 May 4. PMID 33944996
- [Background] Rossetti LZ, Bekheirnia MR, Lewis AM, Mefford HC, Golden-Grant K, Tarczy-Hornoch K, Briere LC, Sweetser DA, Walker MA, Kravets E, Stevenson DA, Bruenner G, Sebastian J, Knapo J, Rosenfeld JA, Marcogliese PC; Undiagnosed Diseases Network; Wangler MF. Missense variants in CTNNB1 can be associated with vitreoretinopathy-Seven new cases of CTNNB1-associated neurodevelopmental disorder including a previously unreported retinal phenotype. Mol Genet Genomic Med. 2021 Jan;9(1):e1542. doi: 10.1002/mgg3.1542. Epub 2020 Dec 22. PMID 33350591
- [Background] Baldridge D, Wangler MF, Bowman AN, Yamamoto S; Undiagnosed Diseases Network; Schedl T, Pak SC, Postlethwait JH, Shin J, Solnica-Krezel L, Bellen HJ, Westerfield M. Model organisms contribute to diagnosis and discovery in the undiagnosed diseases network: current state and a future vision. Orphanet J Rare Dis. 2021 May 7;16(1):206. doi: 10.1186/s13023-021-01839-9. PMID 33962631
- [Background] Wangler MF, Yamamoto S, Chao HT, Posey JE, Westerfield M, Postlethwait J; Members of the Undiagnosed Diseases Network (UDN); Hieter P, Boycott KM, Campeau PM, Bellen HJ. Model Organisms Facilitate Rare Disease Diagnosis and Therapeutic Research. Genetics. 2017 Sep;207(1):9-27. doi: 10.1534/genetics.117.203067. PMID 28874452
- [Background] Harnish JM, Li L, Rogic S, Poirier-Morency G, Kim SY; Undiagnosed Diseases Network; Boycott KM, Wangler MF, Bellen HJ, Hieter P, Pavlidis P, Liu Z, Yamamoto S. ModelMatcher: A scientist-centric online platform to facilitate collaborations between stakeholders of rare and undiagnosed disease research. Hum Mutat. 2022 Jun;43(6):743-759. doi: 10.1002/humu.24364. Epub 2022 Mar 24. PMID 35224820
- [Background] Calame DG, Guo T, Wang C, Garrett L, Jolly A, Dawood M, Kurolap A, Henig NZ, Fatih JM, Herman I, Du H, Mitani T, Becker L, Rathkolb B, Gerlini R, Seisenberger C, Marschall S, Hunter JV, Gerard A, Heidlebaugh A, Challman T, Spillmann RC, Jhangiani SN, Coban-Akdemir Z, Lalani S, Liu L, Revah-Politi A, Iglesias A, Guzman E, Baugh E, Boddaert N, Rondeau S, Ormieres C, Barcia G, Tan QKG, Thiffault I, Pastinen T, Sheikh K, Biliciler S, Mei D, Melani F, Shashi V, Yaron Y, Steele M, Wakeling E, Ostergaard E, Nazaryan-Petersen L; Undiagnosed Diseases Network; Millan F, Santiago-Sim T, Thevenon J, Bruel AL, Thauvin-Robinet C, Popp D, Platzer K, Gawlinski P, Wiszniewski W, Marafi D, Pehlivan D, Posey JE, Gibbs RA, Gailus-Durner V, Guerrini R, Fuchs H, Hrabe de Angelis M, Holter SM, Cheung HH, Gu S, Lupski JR. Monoallelic variation in DHX9, the gene encoding the DExH-box helicase DHX9, underlies neurodevelopment disorders and Charcot-Marie-Tooth disease. Am J Hum Genet. 2023 Aug 3;110(8):1394-1413. doi: 10.1016/j.ajhg.2023.06.013. Epub 2023 Jul 18. PMID 37467750
- [Background] Merselis LC, Jiang SY, Nelson SF, Lee H, Prabaker KK, Baker JL, Munson GP, Butte MJ. MPEG1/Perforin-2 Haploinsufficiency Associated Polymicrobial Skin Infections and Considerations for Interferon-gamma Therapy. Front Immunol. 2020 Nov 3;11:601584. doi: 10.3389/fimmu.2020.601584. eCollection 2020. PMID 33224153
- [Background] Tambe MA, Ng BG, Shimada S, Wolfe LA, Adams DR; Undiagnosed Diseases Network; Gahl WA, Bamshad MJ, Nickerson DA, Malicdan MCV, Freeze HH. Mutations in GET4 disrupt the transmembrane domain recognition complex pathway. J Inherit Metab Dis. 2020 Sep;43(5):1037-1045. doi: 10.1002/jimd.12249. Epub 2020 Jun 3. PMID 32395830
- [Background] Cassini TA, Malicdan MCV, Macnamara EF, Lehky T, Horkayne-Szakaly I, Huang Y, Jones R, Godfrey R, Wolfe L, Gahl WA, Toro C; Undiagnosed Diseases Network. MYH2-associated myopathy caused by a novel splice-site variant. Neuromuscul Disord. 2023 Mar;33(3):257-262. doi: 10.1016/j.nmd.2022.12.014. Epub 2022 Dec 28. PMID 36774715
- [Background] Woods JD, Khanlou N, Lee H, Signer R, Shieh P, Chen J, Herzog M, Palmer C, Martinez-Agosto J; Undiagnosed Diseases Network; Nelson SF. Myopathy associated with homozygous PYROXD1 pathogenic variants detected by genome sequencing. Neuropathology. 2020 Jun;40(3):302-307. doi: 10.1111/neup.12641. Epub 2020 Feb 9. PMID 32037607
- [Background] Wang J, Liu Z, Bellen HJ, Yamamoto S. Navigating MARRVEL, a Web-Based Tool that Integrates Human Genomics and Model Organism Genetics Information. J Vis Exp. 2019 Aug 15;(150):10.3791/59542. doi: 10.3791/59542. PMID 31475990
- [Background] Zhao J, Longo N, Lewis RG, Nicholas TJ, Boyden SE, Andrews A, Larson A; Undiagnosed Diseases Network; Bayrak-Toydemir P, Botto LD, Mao R. Novel molecular mechanism in Malan syndrome uncovered through genome sequencing reanalysis, exon-level Array, and RNA sequencing. Am J Med Genet A. 2024 May;194(5):e63516. doi: 10.1002/ajmg.a.63516. Epub 2024 Jan 2. PMID 38168088
- [Background] Diaz F, Khosa S, Niyazov D, Lee H, Person R, Morrow MM, Signer R, Dorrani N, Zheng A, Herzog M, Freundlich R; Undiagnosed Diseases Network; Birath JB, Cervantes-Manzo Y, Martinez-Agosto JA, Palmer C, Nelson SF, Fogel BL, Mishra SK. Novel NUDT2 variant causes intellectual disability and polyneuropathy. Ann Clin Transl Neurol. 2020 Nov;7(11):2320-2325. doi: 10.1002/acn3.51209. Epub 2020 Oct 15. PMID 33058507
- [Background] Mohanty AK, Vuzman D, Francioli L, Cassa C; Brigham Genomic Medicine; Undiagnosed Diseases Network; Brigham and Women's Hospital FaceBase Project; Toth-Petroczy A, Sunyaev S. novoCaller: a Bayesian network approach for de novo variant calling from pedigree and population sequence data. Bioinformatics. 2019 Apr 1;35(7):1174-1180. doi: 10.1093/bioinformatics/bty749. PMID 30169785
- [Background] Schoch K, McConkie-Rosell A, Walley N, Bhambhani V, Feyma T; Undiagnosed Diseases Network; Pizoli CE, Smith EC, Tan QK, Shashi V. Parental perspectives of episodic irritability in an ultra-rare genetic disorder associated with NACC1. Orphanet J Rare Dis. 2023 Sep 4;18(1):269. doi: 10.1186/s13023-023-02891-3. PMID 37667351
- [Background] Johnson BV, Kumar R, Oishi S, Alexander S, Kasherman M, Vega MS, Ivancevic A, Gardner A, Domingo D, Corbett M, Parnell E, Yoon S, Oh T, Lines M, Lefroy H, Kini U, Van Allen M, Gronborg S, Mercier S, Kury S, Bezieau S, Pasquier L, Raynaud M, Afenjar A, Billette de Villemeur T, Keren B, Desir J, Van Maldergem L, Marangoni M, Dikow N, Koolen DA, VanHasselt PM, Weiss M, Zwijnenburg P, Sa J, Reis CF, Lopez-Otin C, Santiago-Fernandez O, Fernandez-Jaen A, Rauch A, Steindl K, Joset P, Goldstein A, Madan-Khetarpal S, Infante E, Zackai E, Mcdougall C, Narayanan V, Ramsey K, Mercimek-Andrews S, Pena L, Shashi V; Undiagnosed Diseases Network; Schoch K, Sullivan JA, Pinto E Vairo F, Pichurin PN, Ewing SA, Barnett SS, Klee EW, Perry MS, Koenig MK, Keegan CE, Schuette JL, Asher S, Perilla-Young Y, Smith LD, Rosenfeld JA, Bhoj E, Kaplan P, Li D, Oegema R, van Binsbergen E, van der Zwaag B, Smeland MF, Cutcutache I, Page M, Armstrong M, Lin AE, Steeves MA, Hollander ND, Hoffer MJV, Reijnders MRF, Demirdas S, Koboldt DC, Bartholomew D, Mosher TM, Hickey SE, Shieh C, Sanchez-Lara PA, Graham JM Jr, Tezcan K, Schaefer GB, Danylchuk NR, Asamoah A, Jackson KE, Yachelevich N, Au M, Perez-Jurado LA, Kleefstra T, Penzes P, Wood SA, Burne T, Pierson TM, Piper M, Gecz J, Jolly LA. Partial Loss of USP9X Function Leads to a Male Neurodevelopmental and Behavioral Disorder Converging on Transforming Growth Factor beta Signaling. Biol Psychiatry. 2020 Jan 15;87(2):100-112. doi: 10.1016/j.biopsych.2019.05.028. Epub 2019 Jun 29. PMID 31443933
- [Background] Rosenfeld LE, LeBlanc K, Nagy A, Ego BK; Undiagnosed Diseases Network; McCray AT. Participation in a national diagnostic research study: assessing the patient experience. Orphanet J Rare Dis. 2023 Apr 10;18(1):73. doi: 10.1186/s13023-023-02695-5. PMID 37032333
- [Background] Spinelli E, Christensen KR, Bryant E, Schneider A, Rakotomamonjy J, Muir AM, Giannelli J, Littlejohn RO, Roeder ER, Schmidt B, Wilson WG, Marco EJ, Iwama K, Kumada S, Pisano T, Barba C, Vetro A, Brilstra EH, van Jaarsveld RH, Matsumoto N, Goldberg-Stern H, Carney PW, Andrews PI, El Achkar CM, Berkovic S, Rodan LH; Undiagnosed Diseases Network (UDN); McWalter K, Guerrini R, Scheffer IE, Mefford HC, Mandelstam S, Laux L, Millichap JJ, Guemez-Gamboa A, Nairn AC, Carvill GL. Pathogenic MAST3 Variants in the STK Domain Are Associated with Epilepsy. Ann Neurol. 2021 Aug;90(2):274-284. doi: 10.1002/ana.26147. Epub 2021 Jul 13. PMID 34185323
- [Background] Cousin MA, Creighton BA, Breau KA, Spillmann RC, Torti E, Dontu S, Tripathi S, Ajit D, Edwards RJ, Afriyie S, Bay JC, Harper KM, Beltran AA, Munoz LJ, Falcon Rodriguez L, Stankewich MC, Person RE, Si Y, Normand EA, Blevins A, May AS, Bier L, Aggarwal V, Mancini GMS, van Slegtenhorst MA, Cremer K, Becker J, Engels H, Aretz S, MacKenzie JJ, Brilstra E, van Gassen KLI, van Jaarsveld RH, Oegema R, Parsons GM, Mark P, Helbig I, McKeown SE, Stratton R, Cogne B, Isidor B, Cacheiro P, Smedley D, Firth HV, Bierhals T, Kloth K, Weiss D, Fairley C, Shieh JT, Kritzer A, Jayakar P, Kurtz-Nelson E, Bernier RA, Wang T, Eichler EE, van de Laar IMBH, McConkie-Rosell A, McDonald MT, Kemppainen J, Lanpher BC, Schultz-Rogers LE, Gunderson LB, Pichurin PN, Yoon G, Zech M, Jech R, Winkelmann J; Undiagnosed Diseases Network; Genomics England Research Consortium; Beltran AS, Zimmermann MT, Temple B, Moy SS, Klee EW, Tan QK, Lorenzo DN. Pathogenic SPTBN1 variants cause an autosomal dominant neurodevelopmental syndrome. Nat Genet. 2021 Jul;53(7):1006-1021. doi: 10.1038/s41588-021-00886-z. Epub 2021 Jul 1. PMID 34211179
- [Background] Ng BG, Rosenfeld JA, Emrick L, Jain M, Burrage LC, Lee B; Undiagnosed Diseases Network; Craigen WJ, Bearden DR, Graham BH, Freeze HH. Pathogenic Variants in Fucokinase Cause a Congenital Disorder of Glycosylation. Am J Hum Genet. 2018 Dec 6;103(6):1030-1037. doi: 10.1016/j.ajhg.2018.10.021. Epub 2018 Nov 29. PMID 30503518
- [Background] Fountain MD, Oleson DS, Rech ME, Segebrecht L, Hunter JV, McCarthy JM, Lupo PJ, Holtgrewe M, Moran R, Rosenfeld JA, Isidor B, Le Caignec C, Saenz MS, Pedersen RC, Morgan TM, Pfotenhauer JP, Xia F, Bi W, Kang SL, Patel A, Krantz ID, Raible SE, Smith W, Cristian I, Torti E, Juusola J, Millan F, Wentzensen IM, Person RE, Kury S, Bezieau S, Uguen K, Ferec C, Munnich A, van Haelst M, Lichtenbelt KD, van Gassen K, Hagelstrom T, Chawla A, Perry DL, Taft RJ, Jones M, Masser-Frye D, Dyment D, Venkateswaran S, Li C, Escobar LF, Horn D, Spillmann RC, Pena L, Wierzba J, Strom TM, Parenti I, Kaiser FJ, Ehmke N, Schaaf CP. Pathogenic variants in USP7 cause a neurodevelopmental disorder with speech delays, altered behavior, and neurologic anomalies. Genet Med. 2019 Aug;21(8):1797-1807. doi: 10.1038/s41436-019-0433-1. Epub 2019 Jan 25. PMID 30679821
- [Background] McCray AT, LeBlanc K; Undiagnosed Diseases Network. Patients as Partners in Rare Disease Diagnosis and Research. Yale J Biol Med. 2021 Dec 29;94(4):687-692. eCollection 2021 Dec. PMID 34970107
- [Background] Halley MC, Young JL, Fernandez L, Kohler JN; Undiagnosed Diseases Network; Bernstein JA, Wheeler MT, Tabor HK. Perceived utility and disutility of genomic sequencing for pediatric patients: Perspectives from parents with diverse sociodemographic characteristics. Am J Med Genet A. 2022 Apr;188(4):1088-1101. doi: 10.1002/ajmg.a.62619. Epub 2022 Jan 3. PMID 34981646
- [Background] Mukherjee S, Cassini TA, Hu N, Yang T, Li B, Shen W, Moth CW, Rinker DC, Sheehan JH, Cogan JD; Undiagnosed Diseases Network; Newman JH, Hamid R, Macdonald RL, Roden DM, Meiler J, Kuenze G, Phillips JA, Capra JA. Personalized structural biology reveals the molecular mechanisms underlying heterogeneous epileptic phenotypes caused by de novo KCNC2 variants. HGG Adv. 2022 Jul 19;3(4):100131. doi: 10.1016/j.xhgg.2022.100131. eCollection 2022 Oct 13. PMID 36035247
- [Background] Guerrini R, Mei D, Kerti-Szigeti K, Pepe S, Koenig MK, Von Allmen G, Cho MT, McDonald K, Baker J, Bhambhani V, Powis Z, Rodan L, Nabbout R, Barcia G, Rosenfeld JA, Bacino CA, Mignot C, Power LH, Harris CJ, Marjanovic D, Moller RS, Hammer TB; DDD Study; Keski Filppula R, Vieira P, Hildebrandt C, Sacharow S; Undiagnosed Diseases Network; Maragliano L, Benfenati F, Lachlan K, Benneche A, Petit F, de Sainte Agathe JM, Hallinan B, Si Y, Wentzensen IM, Zou F, Narayanan V, Matsumoto N, Boncristiano A, la Marca G, Kato M, Anderson K, Barba C, Sturiale L, Garozzo D, Bei R; ATP6V1A collaborators; Masuelli L, Conti V, Novarino G, Fassio A. Phenotypic and genetic spectrum of ATP6V1A encephalopathy: a disorder of lysosomal homeostasis. Brain. 2022 Aug 27;145(8):2687-2703. doi: 10.1093/brain/awac145. PMID 35675510
- [Background] Bostwick BL, McLean S, Posey JE, Streff HE, Gripp KW, Blesson A, Powell-Hamilton N, Tusi J, Stevenson DA, Farrelly E, Hudgins L, Yang Y, Xia F, Wang X, Liu P, Walkiewicz M, McGuire M, Grange DK, Andrews MV, Hummel M, Madan-Khetarpal S, Infante E, Coban-Akdemir Z, Miszalski-Jamka K, Jefferies JL; Members of the Undiagnosed Diseases Network; Rosenfeld JA, Emrick L, Nugent KM, Lupski JR, Belmont JW, Lee B, Lalani SR. Phenotypic and molecular characterisation of CDK13-related congenital heart defects, dysmorphic facial features and intellectual developmental disorders. Genome Med. 2017 Aug 14;9(1):73. doi: 10.1186/s13073-017-0463-8. PMID 28807008
- [Background] Wang X, Posey JE, Rosenfeld JA, Bacino CA, Scaglia F, Immken L, Harris JM, Hickey SE, Mosher TM, Slavotinek A, Zhang J, Beuten J, Leduc MS, He W, Vetrini F, Walkiewicz MA, Bi W, Xiao R, Liu P, Shao Y, Gezdirici A, Gulec EY, Jiang Y, Darilek SA, Hansen AW, Khayat MM, Pehlivan D, Piard J, Muzny DM, Hanchard N, Belmont JW, Van Maldergem L, Gibbs RA, Eldomery MK, Akdemir ZC, Adesina AM, Chen S, Lee YC; Undiagnosed Diseases Network; Lee B, Lupski JR, Eng CM, Xia F, Yang Y, Graham BH, Moretti P. Phenotypic expansion in DDX3X - a common cause of intellectual disability in females. Ann Clin Transl Neurol. 2018 Sep 15;5(10):1277-1285. doi: 10.1002/acn3.622. eCollection 2018 Oct. PMID 30349862
- [Background] Rodan LH, Spillmann RC, Kurata HT, Lamothe SM, Maghera J, Jamra RA, Alkelai A, Antonarakis SE, Atallah I, Bar-Yosef O, Bilan F, Bjorgo K, Blanc X, Van Bogaert P, Bolkier Y, Burrage LC, Christ BU, Granadillo JL, Dickson P, Donald KA, Dubourg C, Eliyahu A, Emrick L, Engleman K, Gonfiantini MV, Good JM, Kalser J, Kloeckner C, Lachmeijer G, Macchiaiolo M, Nicita F, Odent S, O'Heir E, Ortiz-Gonzalez X, Pacio-Miguez M, Palomares-Bralo M, Pena L, Platzer K, Quinodoz M, Ranza E, Rosenfeld JA, Roulet-Perez E, Santani A, Santos-Simarro F, Pode-Shakked B, Skraban C, Slaugh R, Superti-Furga A, Thiffault I, van Jaabrsveld RH, Vincent M, Wang HG, Zacher P; Undiagnosed Diseases Network; Rush E, Pitt GS, Au PYB, Shashi V. Phenotypic expansion of CACNA1C-associated disorders to include isolated neurological manifestations. Genet Med. 2021 Oct;23(10):1922-1932. doi: 10.1038/s41436-021-01232-8. Epub 2021 Jun 23. PMID 34163037
- [Background] Cassini TA, Robertson AK, Bican AG, Cogan JD, Hannig VL, Newman JH, Hamid R, Phillips JA 3rd; Undiagnosed Diseases Network. Phenotypic heterogeneity of ZMPSTE24 deficiency. Am J Med Genet A. 2018 May;176(5):1175-1179. doi: 10.1002/ajmg.a.38493. Epub 2018 Jan 17. PMID 29341437
- [Background] Castilla-Vallmanya L, Selmer KK, Dimartino C, Rabionet R, Blanco-Sanchez B, Yang S, Reijnders MRF, van Essen AJ, Oufadem M, Vigeland MD, Stadheim B, Houge G, Cox H, Kingston H, Clayton-Smith J, Innis JW, Iascone M, Cereda A, Gabbiadini S, Chung WK, Sanders V, Charrow J, Bryant E, Millichap J, Vitobello A, Thauvin C, Mau-Them FT, Faivre L, Lesca G, Labalme A, Rougeot C, Chatron N, Sanlaville D, Christensen KM, Kirby A, Lewandowski R, Gannaway R, Aly M, Lehman A, Clarke L, Graul-Neumann L, Zweier C, Lessel D, Lozic B, Aukrust I, Peretz R, Stratton R, Smol T, Dieux-Coeslier A, Meira J, Wohler E, Sobreira N, Beaver EM, Heeley J, Briere LC, High FA, Sweetser DA, Walker MA, Keegan CE, Jayakar P, Shinawi M, Kerstjens-Frederikse WS, Earl DL, Siu VM, Reesor E, Yao T, Hegele RA, Vaske OM, Rego S; Undiagnosed Diseases Network, Care4Rare Canada Consortium; Shapiro KA, Wong B, Gambello MJ, McDonald M, Karlowicz D, Colombo R, Serretti A, Pais L, O'Donnell-Luria A, Wray A, Sadedin S, Chong B, Tan TY, Christodoulou J, White SM, Slavotinek A, Barbouth D, Morel Swols D, Parisot M, Bole-Feysot C, Nitschke P, Pingault V, Munnich A, Cho MT, Cormier-Daire V, Balcells S, Lyonnet S, Grinberg D, Amiel J, Urreizti R, Gordon CT. Phenotypic spectrum and transcriptomic profile associated with germline variants in TRAF7. Genet Med. 2020 Jul;22(7):1215-1226. doi: 10.1038/s41436-020-0792-7. Epub 2020 May 7. PMID 32376980
- [Background] Ng BG, Eklund EA, Shiryaev SA, Dong YY, Abbott MA, Asteggiano C, Bamshad MJ, Barr E, Bernstein JA, Chelakkadan S, Christodoulou J, Chung WK, Ciliberto MA, Cousin J, Gardiner F, Ghosh S, Graf WD, Grunewald S, Hammond K, Hauser NS, Hoganson GE, Houck KM, Kohler JN, Morava E, Larson AA, Liu P, Madathil S, McCormack C, Meeks NJL, Miller R, Monaghan KG, Nickerson DA, Palculict TB, Papazoglu GM, Pletcher BA, Scheffer IE, Schenone AB, Schnur RE, Si Y, Rowe LJ, Serrano Russi AH, Russo RS, Thabet F, Tuite A, Villanueva MM, Wang RY, Webster RI, Wilson D, Zalan A; Undiagnosed Diseases Network, University of Washington Center for Mendelian Genomics (UW-CMG); Wolfe LA, Rosenfeld JA, Rhodes L, Freeze HH. Predominant and novel de novo variants in 29 individuals with ALG13 deficiency: Clinical description, biomarker status, biochemical analysis, and treatment suggestions. J Inherit Metab Dis. 2020 Nov;43(6):1333-1348. doi: 10.1002/jimd.12290. Epub 2020 Aug 5. PMID 32681751
- [Background] Sturrock BRH, Macnamara EF, McGuire P, Kruk S, Yang I, Murphy J; Undiagnosed Diseases Network; Tifft CJ, Gordon-Lipkin E. Progressive cerebellar atrophy in a patient with complex II and III deficiency and a novel deleterious variant in SDHA: A Counseling Conundrum. Mol Genet Genomic Med. 2021 Jun;9(6):e1692. doi: 10.1002/mgg3.1692. Epub 2021 May 7. PMID 33960148
- [Background] McConkie-Rosell A, Hooper SR, Pena LDM, Schoch K, Spillmann RC, Jiang YH, Cope H; Undiagnosed Diseases Network; Palmer C, Shashi V. Psychosocial Profiles of Parents of Children with Undiagnosed Diseases: Managing Well or Just Managing? J Genet Couns. 2018 Aug;27(4):935-946. doi: 10.1007/s10897-017-0193-5. Epub 2018 Jan 2. PMID 29297108
- [Background] Han ST, Kim AC, Garcia K, Schimmenti LA, Macnamara E, Network UD, Gahl WA, Malicdan MC, Tifft CJ. PUS7 deficiency in human patients causes profound neurodevelopmental phenotype by dysregulating protein translation. Mol Genet Metab. 2022 Mar;135(3):221-229. doi: 10.1016/j.ymgme.2022.01.103. Epub 2022 Feb 1. PMID 35144859
- [Background] Nil Z, Deshwar AR, Huang Y, Barish S, Zhang X, Choufani S, Le Quesne Stabej P, Hayes I, Yap P, Haldeman-Englert C, Wilson C, Prescott T, Tveten K, Vollo A, Haynes D, Wheeler PG, Zon J, Cytrynbaum C, Jobling R, Blyth M, Banka S, Afenjar A, Mignot C, Robin-Renaldo F, Keren B, Kanca O, Mao X, Wegner DJ, Sisco K, Shinawi M; Undiagnosed Disease Network; Wangler MF, Weksberg R, Yamamoto S, Costain G, Bellen HJ. Rare de novo gain-of-function missense variants in DOT1L are associated with developmental delay and congenital anomalies. Am J Hum Genet. 2023 Nov 2;110(11):1919-1937. doi: 10.1016/j.ajhg.2023.09.009. Epub 2023 Oct 11. PMID 37827158
- [Background] Luo X, Schoch K, Jangam SV, Bhavana VH, Graves HK, Kansagra S, Jasien JM, Stong N, Keren B, Mignot C, Ravelli C; Undiagnosed Diseases Network; Bellen HJ, Wangler MF, Shashi V, Yamamoto S. Rare deleterious de novo missense variants in Rnf2/Ring2 are associated with a neurodevelopmental disorder with unique clinical features. Hum Mol Genet. 2021 Jun 26;30(14):1283-1292. doi: 10.1093/hmg/ddab110. PMID 33864376
- [Background] LeBlanc K, Glanton E, Nagy A, Bater J, Berro T, McGuinness MA, Studwell C; Undiagnosed Diseases Network; Might M. Rare disease patient matchmaking: development and outcomes of an internet case-finding strategy in the Undiagnosed Diseases Network. Orphanet J Rare Dis. 2021 May 10;16(1):210. doi: 10.1186/s13023-021-01825-1. PMID 33971915
- [Background] Kury S, Ebstein F, Molle A, Besnard T, Lee MK, Vignard V, Hery T, Nizon M, Mancini GMS, Giltay JC, Cogne B, McWalter K, Deb W, Mor-Shaked H, Li H, Schnur RE, Wentzensen IM, Denomme-Pichon AS, Fourgeux C, Verheijen FW, Faurie E, Schot R, Stevens CA, Smits DJ, Barr E, Sheffer R, Bernstein JA, Stimach CL, Kovitch E, Shashi V, Schoch K, Smith W, van Jaarsveld RH, Hurst ACE, Smith K, Baugh EH, Bohm SG, Vyhnalkova E, Ryba L, Delnatte C, Neira J, Bonneau D, Toutain A, Rosenfeld JA; Undiagnosed Diseases Network; Audebert-Bellanger S, Gilbert-Dussardier B, Odent S, Laumonnier F, Berger SI, Smith ACM, Bourdeaut F, Stern MH, Redon R, Kruger E, Margueron R, Bezieau S, Poschmann J, Isidor B. Rare germline heterozygous missense variants in BRCA1-associated protein 1, BAP1, cause a syndromic neurodevelopmental disorder. Am J Hum Genet. 2022 Feb 3;109(2):361-372. doi: 10.1016/j.ajhg.2021.12.011. Epub 2022 Jan 19. PMID 35051358
- [Background] Paul MS, Michener SL, Pan H, Pfliger JM, Rosenfeld JA, Lerma VC, Tran A, Longley MA, Lewis RA, Weisz-Hubshman M, Bekheirnia MR, Bekheirnia N, Massingham L, Zech M, Wagner M, Engels H, Cremer K, Mangold E, Peters S, Trautmann J, Mester JL, Guillen Sacoto MJ, Person R, McDonnell PP, Cohen SR, Lusk L, Cohen ASA, Pichon JL, Pastinen T, Zhou D, Engleman K, Racine C, Faivre L, Moutton S, Pichon AD, Schuhmann S, Vasileiou G, Russ-Hall S, Scheffer IE, Carvill GL, Mefford H, Network UD, Bacino CA, Lee BH, Chao HT. Rare variants in PPFIA3 cause delayed development, intellectual disability, autism, and epilepsy. medRxiv [Preprint]. 2023 Mar 29:2023.03.27.23287689. doi: 10.1101/2023.03.27.23287689. PMID 37034625
- [Background] Donkervoort S, Mohassel P, O'Leary M, Bonner DE, Hartley T, Acquaye N, Brull A, Mozaffar T, Saporta MA, Dyment DA, Sampson JB, Pajusalu S, Austin-Tse C, Hurth K, Cohen JS, McWalter K, Warman-Chardon J, Crunk A, Foley AR; Undiagnosed Diseases Network; Mammen AL, Wheeler MT, O'Donnell-Luria A, Bonnemann CG. Recurring homozygous ACTN2 variant (p.Arg506Gly) causes a recessive myopathy. Ann Clin Transl Neurol. 2024 Mar;11(3):629-640. doi: 10.1002/acn3.51983. Epub 2024 Feb 4. PMID 38311799
- [Background] Fazal S, Danzi MC, van Kuilenburg ABP, Reich S, Traschutz A, Bender B, Leen R, Toro C, Usdin K, Hayward B, Adams DR, van Karnebeek CDM, Ferreira CR, D'Sousa P, Network UD, Tekin M, Zuchner S, Synofzik M. Repeat expansions nested within tandem CNVs: a unique structural change in GLS exemplifies the diagnostic challenges of non-coding pathogenic variation. Hum Mol Genet. 2023 Jan 1;32(1):46-54. doi: 10.1093/hmg/ddac173. PMID 35913761
- [Background] Alsentzer E, Finlayson SG, Li MM; Undiagnosed Diseases Network; Kobren SN, Kohane IS. Simulation of undiagnosed patients with novel genetic conditions. Nat Commun. 2023 Oct 12;14(1):6403. doi: 10.1038/s41467-023-41980-6. PMID 37828001
- [Background] Ng BG, Sosicka P, Agadi S, Almannai M, Bacino CA, Barone R, Botto LD, Burton JE, Carlston C, Chung BH, Cohen JS, Coman D, Dipple KM, Dorrani N, Dobyns WB, Elias AF, Epstein L, Gahl WA, Garozzo D, Hammer TB, Haven J, Heron D, Herzog M, Hoganson GE, Hunter JM, Jain M, Juusola J, Lakhani S, Lee H, Lee J, Lewis K, Longo N, Lourenco CM, Mak CCY, McKnight D, Mendelsohn BA, Mignot C, Mirzaa G, Mitchell W, Muhle H, Nelson SF, Olczak M, Palmer CGS, Partikian A, Patterson MC, Pierson TM, Quinonez SC, Regan BM, Ross ME, Guillen Sacoto MJ, Scaglia F, Scheffer IE, Segal D, Singhal NS, Striano P, Sturiale L, Symonds JD, Tang S, Vilain E, Willis M, Wolfe LA, Yang H, Yano S, Powis Z, Suchy SF, Rosenfeld JA, Edmondson AC, Grunewald S, Freeze HH. SLC35A2-CDG: Functional characterization, expanded molecular, clinical, and biochemical phenotypes of 30 unreported Individuals. Hum Mutat. 2019 Jul;40(7):908-925. doi: 10.1002/humu.23731. Epub 2019 Apr 24. PMID 30817854
- [Background] Beck DB, Ferrada MA, Sikora KA, Ombrello AK, Collins JC, Pei W, Balanda N, Ross DL, Ospina Cardona D, Wu Z, Patel B, Manthiram K, Groarke EM, Gutierrez-Rodrigues F, Hoffmann P, Rosenzweig S, Nakabo S, Dillon LW, Hourigan CS, Tsai WL, Gupta S, Carmona-Rivera C, Asmar AJ, Xu L, Oda H, Goodspeed W, Barron KS, Nehrebecky M, Jones A, Laird RS, Deuitch N, Rowczenio D, Rominger E, Wells KV, Lee CR, Wang W, Trick M, Mullikin J, Wigerblad G, Brooks S, Dell'Orso S, Deng Z, Chae JJ, Dulau-Florea A, Malicdan MCV, Novacic D, Colbert RA, Kaplan MJ, Gadina M, Savic S, Lachmann HJ, Abu-Asab M, Solomon BD, Retterer K, Gahl WA, Burgess SM, Aksentijevich I, Young NS, Calvo KR, Werner A, Kastner DL, Grayson PC. Somatic Mutations in UBA1 and Severe Adult-Onset Autoinflammatory Disease. N Engl J Med. 2020 Dec 31;383(27):2628-2638. doi: 10.1056/NEJMoa2026834. Epub 2020 Oct 27. PMID 33108101
- [Background] Kelly M, Park M, Mihalek I, Rochtus A, Gramm M, Perez-Palma E, Axeen ET, Hung CY, Olson H, Swanson L, Anselm I, Briere LC, High FA, Sweetser DA; Undiagnosed Diseases Network; Kayani S, Snyder M, Calvert S, Scheffer IE, Yang E, Waugh JL, Lal D, Bodamer O, Poduri A. Spectrum of neurodevelopmental disease associated with the GNAO1 guanosine triphosphate-binding region. Epilepsia. 2019 Mar;60(3):406-418. doi: 10.1111/epi.14653. Epub 2019 Jan 25. PMID 30682224
- [Background] Srivastava S, Shaked HM, Gable K, Gupta SD, Pan X, Somashekarappa N, Han G, Mohassel P, Gotkine M, Doney E, Goldenberg P, Tan QKG, Gong Y, Kleinstiver B, Wishart B, Cope H, Pires CB, Stutzman H, Spillmann RC; Undiagnosed Disease Network; Sadjadi R, Elpeleg O, Lee CH, Bellen HJ, Edvardson S, Eichler F, Dunn TM. SPTSSA variants alter sphingolipid synthesis and cause a complex hereditary spastic paraplegia. Brain. 2023 Apr 19;146(4):1420-1435. doi: 10.1093/brain/awac460. PMID 36718090
- [Background] Webb-Robertson BM, Stratton KG, Kyle JE, Kim YM, Bramer LM, Waters KM, Koeller DM, Metz TO. Statistically Driven Metabolite and Lipid Profiling of Patients from the Undiagnosed Diseases Network. Anal Chem. 2020 Jan 21;92(2):1796-1803. doi: 10.1021/acs.analchem.9b03522. Epub 2019 Dec 5. PMID 31742994
- [Background] DeFilippis EM, Solomon M, Loscalzo J. Superior Mesenteric Artery Dissection: Classical Presentation, Novel Genetic Determinants. JACC Case Rep. 2021 Feb 24;3(4):690-693. doi: 10.1016/j.jaccas.2020.12.034. eCollection 2021 Apr. PMID 34317605
- [Background] Vollger MR, Korlach J, Eldred KC, Swanson E, Underwood JG, Cheng YH, Ranchalis J, Mao Y, Blue EE, Schwarze U, Munson KM, Saunders CT, Wenger AM, Allworth A, Chanprasert S, Duerden BL, Glass I, Horike-Pyne M, Kim M, Leppig KA, McLaughlin IJ, Ogawa J, Rosenthal EA, Sheppeard S, Sherman SM, Strohbehn S, Yuen AL; University of Washington Center for Mendelian Genomics (UW-CMG), Undiagnosed Diseases Network (UDN); Reh TA, Byers PH, Bamshad MJ, Hisama FM, Jarvik GP, Sancak Y, Dipple KM, Stergachis AB. Synchronized long-read genome, methylome, epigenome, and transcriptome for resolving a Mendelian condition. bioRxiv [Preprint]. 2023 Sep 27:2023.09.26.559521. doi: 10.1101/2023.09.26.559521. PMID 37808736
- [Background] Forsyth R, Parisi MA, Altintas B, Malicdan MC, Vilboux T, Knoll J, Brooks BP, Zein WM, Gahl WA, Toro C, Gunay-Aygun M. Systematic analysis of physical examination characteristics of 94 individuals with Joubert syndrome: Keys to suspecting the diagnosis. Am J Med Genet C Semin Med Genet. 2022 Mar;190(1):121-130. doi: 10.1002/ajmg.c.31966. Epub 2022 Mar 21. PMID 35312150
- [Background] Bellen HJ, Wangler MF, Yamamoto S. The fruit fly at the interface of diagnosis and pathogenic mechanisms of rare and common human diseases. Hum Mol Genet. 2019 Nov 21;28(R2):R207-R214. doi: 10.1093/hmg/ddz135. PMID 31227826
- [Background] Senderek J, Lassuthova P, Kabzinska D, Abreu L, Baets J, Beetz C, Braathen GJ, Brenner D, Dalton J, Dankwa L, Deconinck T, De Jonghe P, Drager B, Eggermann K, Ellis M, Fischer C, Stojkovic T, Herrmann DN, Horvath R, Hoyer H, Iglseder S, Kennerson M, Kinslechner K, Kohler JN, Kurth I, Laing NG, Lamont PJ, Wolfgang N L, Ludolph A, Marques W Jr, Nicholson G, Ong R, Petri S, Ravenscroft G, Rebelo A, Ricci G, Rudnik-Schoneborn S, Schirmacher A, Schlotter-Weigel B, Schoels L, Schule R, Synofzik M, Francou B, Strom TM, Wagner J, Walk D, Wanschitz J, Weinmann D, Weishaupt J, Wiessner M, Windhager R, Young P, Zuchner S, Toegel S, Seeman P, Kochanski A, Auer-Grumbach M. The genetic landscape of axonal neuropathies in the middle-aged and elderly: Focus on MME. Neurology. 2020 Dec 15;95(24):e3163-e3179. doi: 10.1212/WNL.0000000000011132. Epub 2020 Nov 3. PMID 33144514
- [Background] McConkie-Rosell A, Schoch K, Sullivan J, Cope H, Spillmann R, Palmer CGS, Pena L, Jiang YH, Daniels N, Walley N, Tan KG; Undiagnosed Diseases Network; Hooper SR, Shashi V. The genome empowerment scale: An assessment of parental empowerment in families with undiagnosed disease. Clin Genet. 2019 Dec;96(6):521-531. doi: 10.1111/cge.13635. Epub 2019 Oct 8. PMID 31448412
- [Background] Barish S, Senturk M, Schoch K, Minogue AL, Lopergolo D, Fallerini C, Harland J, Seemann JH, Stong N, Kranz PG, Kansagra S, Mikati MA, Jasien J, El-Dairi M, Galluzzi P; Undiagnosed Diseases Network; Ariani F, Renieri A, Mari F, Wangler MF, Arur S, Jiang YH, Yamamoto S, Shashi V, Bellen HJ. The microRNA processor DROSHA is a candidate gene for a severe progressive neurological disorder. Hum Mol Genet. 2022 Aug 25;31(17):2934-2950. doi: 10.1093/hmg/ddac085. PMID 35405010
- [Background] Gahl WA, Mulvihill JJ, Toro C, Markello TC, Wise AL, Ramoni RB, Adams DR, Tifft CJ; UDN. The NIH Undiagnosed Diseases Program and Network: Applications to modern medicine. Mol Genet Metab. 2016 Apr;117(4):393-400. doi: 10.1016/j.ymgme.2016.01.007. Epub 2016 Jan 22. PMID 26846157
- [Background] Huang Y, Lemire G, Briere LC, Liu F, Wessels MW, Wang X, Osmond M, Kanca O, Lu S, High FA, Walker MA, Rodan LH; Undiagnosed Diseases Network; Care4Rare Canada Consortium; Kernohan KD, Sweetser DA, Boycott KM, Bellen HJ. The recurrent de novo c.2011C>T missense variant in MTSS2 causes syndromic intellectual disability. Am J Hum Genet. 2022 Oct 6;109(10):1923-1931. doi: 10.1016/j.ajhg.2022.08.011. Epub 2022 Sep 5. PMID 36067766
- [Background] Aday AW, Krier JB, Pallais JC, Fieg EL, MacRae CA, Loscalzo J; Members of the UDN. The Undiagnosed Diseases Network as a Tool for Graduate Medical Education. Am J Med. 2020 Feb;133(2):e18-e22. doi: 10.1016/j.amjmed.2019.06.034. Epub 2019 Jul 10. No abstract available. PMID 31301294
- [Background] Ramoni RB, Mulvihill JJ, Adams DR, Allard P, Ashley EA, Bernstein JA, Gahl WA, Hamid R, Loscalzo J, McCray AT, Shashi V, Tifft CJ; Undiagnosed Diseases Network; Wise AL. The Undiagnosed Diseases Network: Accelerating Discovery about Health and Disease. Am J Hum Genet. 2017 Feb 2;100(2):185-192. doi: 10.1016/j.ajhg.2017.01.006. PMID 28157539
- [Background] Macnamara EF, D'Souza P; Undiagnosed Diseases Network; Tifft CJ. The undiagnosed diseases program: Approach to diagnosis. Transl Sci Rare Dis. 2020 Apr 13;4(3-4):179-188. doi: 10.3233/TRD-190045. PMID 32477883
- [Background] Akula SK, Marciano JH, Lim Y, Exposito-Alonso D, Hylton NK, Hwang GH, Neil JE, Dominado N, Bunton-Stasyshyn RK, Song JHT, Talukdar M, Schmid A, Teboul L, Mo A, Shin T, Finander B, Beck SG, Yeh RC, Otani A, Qian X, DeGennaro EM, Alkuraya FS, Maddirevula S, Cascino GD, Giannini C; Undiagnosed Diseases Network; Burrage LC, Rosenfield JA, Ketkar S, Clark GD, Bacino C, Lewis RA, Segal RA, Bazan JF, Smith KA, Golden JA, Cho G, Walsh CA. TMEM161B regulates cerebral cortical gyration, Sonic Hedgehog signaling, and ciliary structure in the developing central nervous system. Proc Natl Acad Sci U S A. 2023 Jan 24;120(4):e2209964120. doi: 10.1073/pnas.2209964120. Epub 2023 Jan 20. PMID 36669111
- [Background] Goodman LD, Cope H, Nil Z, Ravenscroft TA, Charng WL, Lu S, Tien AC, Pfundt R, Koolen DA, Haaxma CA, Veenstra-Knol HE, Wassink-Ruiter JSK, Wevers MR, Jones M, Walsh LE, Klee VH, Theunis M, Legius E, Steel D, Barwick KES, Kurian MA, Mohammad SS, Dale RC, Terhal PA, van Binsbergen E, Kirmse B, Robinette B, Cogne B, Isidor B, Grebe TA, Kulch P, Hainline BE, Sapp K, Morava E, Klee EW, Macke EL, Trapane P, Spencer C, Si Y, Begtrup A, Moulton MJ, Dutta D, Kanca O; Undiagnosed Diseases Network; Wangler MF, Yamamoto S, Bellen HJ, Tan QK. TNPO2 variants associate with human developmental delays, neurologic deficits, and dysmorphic features and alter TNPO2 activity in Drosophila. Am J Hum Genet. 2021 Sep 2;108(9):1669-1691. doi: 10.1016/j.ajhg.2021.06.019. Epub 2021 Jul 26. PMID 34314705
- [Background] Murdock DR, Dai H, Burrage LC, Rosenfeld JA, Ketkar S, Muller MF, Yepez VA, Gagneur J, Liu P, Chen S, Jain M, Zapata G, Bacino CA, Chao HT, Moretti P, Craigen WJ, Hanchard NA; Undiagnosed Diseases Network; Lee B. Transcriptome-directed analysis for Mendelian disease diagnosis overcomes limitations of conventional genomic testing. J Clin Invest. 2021 Jan 4;131(1):e141500. doi: 10.1172/JCI141500. PMID 33001864
- [Background] Gu S, Chen CA, Rosenfeld JA, Cope H, Launay N, Flanigan KM, Waldrop MA, Schrader R, Juusola J, Goker-Alpan O, Milunsky A, Schluter A, Troncoso M, Pujol A, Tan QK, Schaaf CP, Meng L. Truncating variants in UBAP1 associated with childhood-onset nonsyndromic hereditary spastic paraplegia. Hum Mutat. 2020 Mar;41(3):632-640. doi: 10.1002/humu.23950. Epub 2019 Nov 25. PMID 31696996
- [Background] Bowles B, Ferrer A, Nishimura CJ, Pinto E Vairo F, Rey T, Leheup B, Sullivan J, Schoch K, Stong N, Agolini E, Cocciadiferro D, Williams A, Cummings A, Loddo S, Genovese S, Roadhouse C, McWalter K; Undiagnosed Diseases Network; Wentzensen IM, Li C, Babovic-Vuksanovic D, Lanpher BC, Dentici ML, Ankala A, Hamm JA, Dallapiccola B, Radio FC, Shashi V, Gerard B, Bloch-Zupan A, Smith RJ, Klee EW. TSPEAR variants are primarily associated with ectodermal dysplasia and tooth agenesis but not hearing loss: A novel cohort study. Am J Med Genet A. 2021 Aug;185(8):2417-2433. doi: 10.1002/ajmg.a.62347. Epub 2021 May 27. PMID 34042254
- [Background] Palmer CGS, McConkie-Rosell A, Holm IA, LeBlanc K, Sinsheimer JS, Briere LC, Dorrani N, Herzog MR, Lincoln S, Schoch K, Spillmann RC, Brokamp E; Undiagnosed Diseases Network. Understanding Adult Participant and Parent Empowerment Prior to Evaluation in the Undiagnosed Diseases Network. J Genet Couns. 2018 Sep;27(5):1087-1101. doi: 10.1007/s10897-018-0228-6. Epub 2018 Mar 1. PMID 29497923
- [Background] Taruscio D, Salvatore M, Lumaka A, Carta C, Cellai LL, Ferrari G, Sciascia S, Groft S, Alanay Y, Azam M, Baynam G, Cederroth H, Cutiongco-de la Paz EM, Dissanayake VHW, Giugliani R, Gonzaga-Jauregui C, Hettiarachchi D, Kvlividze O, Landoure G, Makay P, Melegh B, Ozbek U, Puri RD, Romero V, Scaria V, Jamuar SS, Shotelersuk V, Roccatello D, Gahl WA, Wiafe SA, Bodamer O, Posada M. Undiagnosed diseases: Needs and opportunities in 20 countries participating in the Undiagnosed Diseases Network International. Front Public Health. 2023 Mar 2;11:1079601. doi: 10.3389/fpubh.2023.1079601. eCollection 2023. PMID 36935719
- [Background] Sciascia S, Roccatello D, Salvatore M, Carta C, Cellai LL, Ferrari G, Lumaka A, Groft S, Alanay Y, Azam M, Baynam G, Cederroth H, Cutiongco-de la Paz EM, Dissanayake VHW, Giugliani R, Gonzaga-Jauregui C, Hettiarachchi D, Kvlividze O, Landoure G, Makay P, Melegh B, Ozbek U, Puri RD, Romero VI, Scaria V, Jamuar SS, Shotelersuk V, Gahl WA, Wiafe SA, Bodamer O, Posada M, Taruscio D. Unmet needs in countries participating in the undiagnosed diseases network international: an international survey considering national health care and economic indicators. Front Public Health. 2023 Sep 26;11:1248260. doi: 10.3389/fpubh.2023.1248260. eCollection 2023. PMID 37822540
- [Background] McConkie-Rosell A, Spillmann RC, Schoch K, Sullivan JA, Walley N, McDonald M; Undiagnosed Diseases Network; Hooper SR, Shashi V. Unraveling non-participation in genomic research: A complex interplay of barriers, facilitators, and sociocultural factors. J Genet Couns. 2023 Oct;32(5):993-1008. doi: 10.1002/jgc4.1707. Epub 2023 Apr 2. PMID 37005744
- [Background] Wang J, Mao D, Fazal F, Kim SY, Yamamoto S, Bellen H, Liu Z. Using MARRVEL v1.2 for Bioinformatics Analysis of Human Genes and Variant Pathogenicity. Curr Protoc Bioinformatics. 2019 Sep;67(1):e85. doi: 10.1002/cpbi.85. PMID 31524990
- [Background] Scala M, Nishikawa M, Ito H, Tabata H, Khan T, Accogli A, Davids L, Ruiz A, Chiurazzi P, Cericola G, Schulte B, Monaghan KG, Begtrup A, Torella A, Pinelli M, Denomme-Pichon AS, Vitobello A, Racine C, Mancardi MM, Kiss C, Guerin A, Wu W, Gabau Vila E, Mak BC, Martinez-Agosto JA, Gorin MB, Duz B, Bayram Y, Carvalho CMB, Vengoechea JE, Chitayat D, Tan TY, Callewaert B, Kruse B, Bird LM, Faivre L, Zollino M, Biskup S; Undiagnosed Diseases Network; Telethon Undiagnosed Diseases Program; Striano P, Nigro V, Severino M, Capra V, Costain G, Nagata KI. Variant-specific changes in RAC3 function disrupt corticogenesis in neurodevelopmental phenotypes. Brain. 2022 Sep 14;145(9):3308-3327. doi: 10.1093/brain/awac106. PMID 35851598
- [Background] Marbach F, Stoyanov G, Erger F, Stratakis CA, Settas N, London E, Rosenfeld JA, Torti E, Haldeman-Englert C, Sklirou E, Kessler E, Ceulemans S, Nelson SF, Martinez-Agosto JA, Palmer CGS, Signer RH; Undiagnosed Diseases Network; Andrews MV, Grange DK, Willaert R, Person R, Telegrafi A, Sievers A, Laugsch M, Theiss S, Cheng Y, Lichtarge O, Katsonis P, Stocco A, Schaaf CP. Variants in PRKAR1B cause a neurodevelopmental disorder with autism spectrum disorder, apraxia, and insensitivity to pain. Genet Med. 2021 Aug;23(8):1465-1473. doi: 10.1038/s41436-021-01152-7. Epub 2021 Apr 8. PMID 33833410
- [Background] Holt JM, Wilk B, Birch CL, Brown DM, Gajapathy M, Moss AC, Sosonkina N, Wilk MA, Anderson JA, Harris JM, Kelly JM, Shaterferdosian F, Uno-Antonison AE, Weborg A; Undiagnosed Diseases Network; Worthey EA. VarSight: prioritizing clinically reported variants with binary classification algorithms. BMC Bioinformatics. 2019 Oct 15;20(1):496. doi: 10.1186/s12859-019-3026-8. PMID 31615419
- [Background] Murdock DR, Rosenfeld JA, Lee B. What Has the Undiagnosed Diseases Network Taught Us About the Clinical Applications of Genomic Testing? Annu Rev Med. 2022 Jan 27;73:575-585. doi: 10.1146/annurev-med-042120-014904. PMID 35084988
- [Background] Cassini TA, Duncan L, Rives LC, Newman JH, Phillips JA, Koziura ME, Brault J, Hamid R, Cogan J; Undiagnosed Diseases Network. Whole genome sequencing reveals novel IGHMBP2 variant leading to unique cryptic splice-site and Charcot-Marie-Tooth phenotype with early onset symptoms. Mol Genet Genomic Med. 2019 Jun;7(6):e00676. doi: 10.1002/mgg3.676. Epub 2019 Apr 25. PMID 31020813
- [Background] King KA, Wegner DJ, Bucelli RC, Shapiro J, Paul AJ, Dickson PI, Wambach JA; Undiagnosed Disease Network (UDN). Whole-Genome and Long-Read Sequencing Identify a Novel Mechanism in RFC1 Resulting in CANVAS Syndrome. Neurol Genet. 2022 Nov 1;8(6):e200036. doi: 10.1212/NXG.0000000000200036. eCollection 2022 Dec. PMID 36524104
- [Background] Keehan L, Haviland I, Gofin Y, Swanson LC, El Achkar CM, Schreiber J, VanNoy GE, O'Heir E, O'Donnell-Luria A, Lewis RA, Magoulas P, Tran A, Azamian MS, Chao HT, Pham L, Samaco RC, Elsea S, Thorpe E, Kesari A, Perry D, Lee B, Lalani SR, Rosenfeld JA, Olson HE, Burrage LC; Undiagnosed Diseases Network. Wide range of phenotypic severity in individuals with late truncations unique to the predominant CDKL5 transcript in the brain. Am J Med Genet A. 2022 Dec;188(12):3516-3524. doi: 10.1002/ajmg.a.62940. Epub 2022 Aug 7. PMID 35934918
- [Background] Reuter CM, Kohler JN, Bonner D, Zastrow D, Fernandez L, Dries A, Marwaha S, Davidson J, Brokamp E, Herzog M, Hong J, Macnamara E, Rosenfeld JA, Schoch K, Spillmann R; Undiagnosed Diseases Network; Loscalzo J, Krier J, Stoler J, Sweetser D, Palmer CGS, Phillips JA, Shashi V, Adams DA, Yang Y, Ashley EA, Fisher PG, Mulvihill JJ, Bernstein JA, Wheeler MT. Yield of whole exome sequencing in undiagnosed patients facing insurance coverage barriers to genetic testing. J Genet Couns. 2019 Dec;28(6):1107-1118. doi: 10.1002/jgc4.1161. Epub 2019 Sep 3. PMID 31478310
- [Background] Blanco-Sanchez B, Clement A, Stednitz SJ, Kyle J, Peirce JL, McFadden M, Wegner J, Phillips JB, Macnamara E, Huang Y, Adams DR, Toro C, Gahl WA, Malicdan MCV, Tifft CJ, Zink EM, Bloodsworth KJ, Stratton KG; Undiagnosed Diseases Network; Koeller DM, Metz TO, Washbourne P, Westerfield M. yippee like 3 (ypel3) is a novel gene required for myelinating and perineurial glia development. PLoS Genet. 2020 Jun 16;16(6):e1008841. doi: 10.1371/journal.pgen.1008841. eCollection 2020 Jun. PMID 32544203
- [Background] Peretz RH, Zein WM, Hufnagel RB, Ku C, Godfrey R, Wolfe L, Adams D, Gahl W, Toro C. A de novo hexokinase 1 (HK1) variant presenting as Boucher-Neuhauser syndrome. Am J Med Genet A. 2023 Feb;191(2):624-629. doi: 10.1002/ajmg.a.63045. Epub 2022 Dec 21. PMID 36541585
- [Background] Dutta D, Kanca O, Byeon SK, Marcogliese PC, Zuo Z, Shridharan RV, Park JH; Undiagnosed Diseases Network; Lin G, Ge M, Heimer G, Kohler JN, Wheeler MT, Kaipparettu BA, Pandey A, Bellen HJ. A defect in mitochondrial fatty acid synthesis impairs iron metabolism and causes elevated ceramide levels. Nat Metab. 2023 Sep;5(9):1595-1614. doi: 10.1038/s42255-023-00873-0. Epub 2023 Aug 31. PMID 37653044
- [Background] Furuta Y, Nelson ET, Neumann SM, Phillips JA 3rd, Hamid R, Tinker RJ, Cogan JD, Rives L, Newman JH; Undiagnosed Diseases Network. A medical odyssey of a 72-year-old man with Charcot-Marie-Tooth disease type 2 newly diagnosed with biallelic variants in SORD gene causing sorbitol dehydrogenase deficiency. Am J Med Genet A. 2023 Dec;191(12):2873-2877. doi: 10.1002/ajmg.a.63383. Epub 2023 Aug 25. PMID 37622199
- [Background] Bouzinier MA, Etin D, Trifonov SI, Evdokimova VN, Ulitin V, Shen J, Kokorev A, Ghazani AA, Chekaluk Y, Albertyn Z, Giersch A, Morton CC, Abraamyan F, Bendapudi PK, Sunyaev S, Undiagnosed Diseases Network, Brigham Genomic Medicine, SEQuencing A Baby For An Optimal Outcome, Quantori, Krier JB. AnFiSA: An open-source computational platform for the analysis of sequencing data for rare genetic disease. J Biomed Inform. 2022 Sep;133:104174. doi: 10.1016/j.jbi.2022.104174. Epub 2022 Aug 23. PMID 35998814
- [Background] Peart LS, Gonzalez J, Bivona S, Latchman K, Torres L; Undiagnosed Diagnosis Network; Tekin M. Bilateral choanal stenosis in auriculocondylar syndrome caused by a PLCB4 variant. Am J Med Genet A. 2022 Apr;188(4):1307-1310. doi: 10.1002/ajmg.a.62634. Epub 2022 Jan 7. PMID 34995019
- [Background] Kimera L, Nadimpalli S, Kurup S, Cole FS, Huang R, Sisco K, Ranaivo HR, Shinawi M, Dickson P, Mian A, Reynolds M, Undiagnosed Diseases Network. Case report: ocular manifestations of a gain-of-function mutation in CLCN6, a newly diagnosed disease. Ophthalmic Genet. 2024 Jun;45(3):271-274. doi: 10.1080/13816810.2023.2291683. Epub 2023 Dec 14. PMID 38095064
- [Background] Ward SK, Wadley A, Tsai CA, Benke PJ, Emrick L, Fisher K, Houck KM, Dai H; Undiagnosed Diseases Network; Guillen Sacoto MJ, Craigen W, Glaser K, Murdock DR, Rohena L, Diderich KEM, Bruggenwirth HT, Lee B, Bacino C, Burrage LC, Rosenfeld JA. De novo missense variants in ZBTB47 are associated with developmental delays, hypotonia, seizures, gait abnormalities, and variable movement abnormalities. Am J Med Genet A. 2024 Jan;194(1):17-30. doi: 10.1002/ajmg.a.63399. Epub 2023 Sep 25. PMID 37743782
- [Background] Andrews JC, Mok JW, Kanca O, Jangam S, Tifft C, Macnamara EF, Russell BE, Wang LK; Undiagnosed Diseases Network; Nelson SF, Bellen HJ, Yamamoto S, Malicdan MCV, Wangler MF. De novo variants in MRTFB have gain-of-function activity in Drosophila and are associated with a novel neurodevelopmental phenotype with dysmorphic features. Genet Med. 2023 Jun;25(6):100833. doi: 10.1016/j.gim.2023.100833. Epub 2023 Mar 31. PMID 37013900
- [Background] Montano C, Cassini T, Ziegler SG, Boehm M, Nicoli ER, Mindell JA, Soldatos AG, Manoli I, Wolfe L, Macnamara EF, Malicdan MCV, Adams DR, Tifft CJ, Toro C, Gahl WA. Diagnosis and discovery: Insights from the NIH Undiagnosed Diseases Program. J Inherit Metab Dis. 2022 Sep;45(5):907-918. doi: 10.1002/jimd.12506. Epub 2022 May 16. PMID 35490291
- [Background] Mohajeri A, Vaseghi-Shanjani M, Rosenfeld JA, Yang GX, Lu H, Sharma M, Lin S, Salman A, Waqas M, Sababi Azamian M, Worley KC, Del Bel KL, Kozak FK, Rahmanian R, Biggs CM, Hildebrand KJ, Lalani SR, Nicholas SK, Scott DA, Mostafavi S, van Karnebeek C, Henkelman E, Halparin J, Yang CL, Armstrong L; Undiagnosed Diseases Network; Care4Rare Canada Consortium; Turvey SE, Lehman A. Dominant negative variants in IKZF2 cause ICHAD syndrome, a new disorder characterised by immunodysregulation, craniofacial anomalies, hearing impairment, athelia and developmental delay. J Med Genet. 2023 Nov;60(11):1092-1104. doi: 10.1136/jmg-2022-109127. Epub 2023 Jun 14. PMID 37316189
- [Background] Chong SC, Cao Y, Fung ELW, Kleppe S, Gripp KW, Hertecant J, El-Hattab AW, Suleiman J, Clark G, von Allmen G, Rodziyevska O, Lewis RA, Rosenfeld JA, Dong J; Undiagnosed Diseases Network; Wang X, Miller MJ, Bi W, Liu P, Scaglia F. Expansion of the clinical and molecular spectrum of WWOX-related epileptic encephalopathy. Am J Med Genet A. 2023 Mar;191(3):776-785. doi: 10.1002/ajmg.a.63074. Epub 2022 Dec 19. PMID 36537114
- [Background] Chen YH, Zastrow DB, Metcalfe RD, Gartner L, Krause F, Morton CJ, Marwaha S, Fresard L, Huang Y, Zhao C, McCormack C, Bick D, Worthey EA, Eng CM, Gold J, Undiagnosed Diseases Network, Montgomery SB, Fisher PG, Ashley EA, Wheeler MT, Parker MW, Shanmugasundaram V, Putoczki TL, Schmidt-Arras D, Laurence A, Bernstein JA, Griffin MDW, Uhlig HH. Functional and structural analysis of cytokine-selective IL6ST defects that cause recessive hyper-IgE syndrome. J Allergy Clin Immunol. 2021 Aug;148(2):585-598. doi: 10.1016/j.jaci.2021.02.044. Epub 2021 Mar 23. PMID 33771552
- [Background] Weixel T, Wolfe L, Macnamara EF. Genetic counseling for congenital disorders of glycosylation (CDG). J Genet Couns. 2024 Dec;33(6):1358-1364. doi: 10.1002/jgc4.1856. Epub 2024 Jan 19. PMID 38240170
- [Background] Kohler JN, Glanton E, Boyd BM, Sillari CH, Marwaha S; Undiagnosed Diseases Network; Wheeler MT. Genetic counselor roles in the undiagnosed diseases network research study: Clinical care, collaboration, and curation. J Genet Couns. 2022 Apr;31(2):326-337. doi: 10.1002/jgc4.1493. Epub 2021 Aug 10. PMID 34374469
- [Background] Geng LN, Kohler JN, Levonian P; Members of the Undiagnosed Diseases Network; Bernstein JA, Ford JM, Ahuja N, Witteles R, Hom J, Wheeler M. Genomics in medicine: a novel elective rotation for internal medicine residents. Postgrad Med J. 2019 Oct;95(1128):569-572. doi: 10.1136/postgradmedj-2018-136355. Epub 2019 Aug 22. PMID 31439813
- [Background] Rosenfeld JA, Xiao R, Bekheirnia MR, Kanani F, Parker MJ, Koenig MK, van Haeringen A, Ruivenkamp C, Rosmaninho-Salgado J, Almeida PM, Sa J, Pinto Basto J, Palen E, Oetjens KF, Burrage LC, Xia F, Liu P, Eng CM; Undiagnosed Diseases Network; Yang Y, Posey JE, Lee BH. Heterozygous variants in SPTBN1 cause intellectual disability and autism. Am J Med Genet A. 2021 Jul;185(7):2037-2045. doi: 10.1002/ajmg.a.62201. Epub 2021 Apr 13. PMID 33847457
- [Background] Yoo B, Birgmeier J, Bernstein JA, Bejerano G. InpherNet accelerates monogenic disease diagnosis using patients' candidate genes' neighbors. Genet Med. 2021 Oct;23(10):1984-1992. doi: 10.1038/s41436-021-01238-2. Epub 2021 Jul 6. PMID 34230641
- [Background] Brokamp E, Koziura ME, Phillips JA 3rd, Tang LA, Cogan JD, Rives LC, Robertson AK, Duncan L, Bican A, Peterson JF, Newman JH, Hamid R, Bastarache L; Undiagnosed Diseases Network. One is the loneliest number: genotypic matchmaking using the electronic health record. Genet Med. 2021 Oct;23(10):1830-1832. doi: 10.1038/s41436-021-01179-w. Epub 2021 Jul 6. No abstract available. PMID 34230636
- [Background] Panneerselvam S, Wang J, Zhu W, Dai H, Pappas JG, Rabin R, Low KJ, Rosenfeld JA, Emrick L, Xiao R, Xia F, Yang Y, Eng CM, Anderson A, Chau V, Soler-Alfonso C, Streff H, Lalani SR, Mercimek-Andrews S; Undiagnosed Diseases Network; DDD Study; Bi W. PPP3CA truncating variants clustered in the regulatory domain cause early-onset refractory epilepsy. Clin Genet. 2021 Aug;100(2):227-233. doi: 10.1111/cge.13979. Epub 2021 Jun 1. PMID 33963760
- [Background] Furuta Y, Tinker RJ, Gulsevin A, Neumann SM, Hamid R, Cogan JD, Rives L, Liu Q, Chen HC, Joos KM, Phillips JA 3rd; Undiagnosed Diseases Network. Probable digenic inheritance of Diamond-Blackfan anemia. Am J Med Genet A. 2024 Mar;194(3):e63454. doi: 10.1002/ajmg.a.63454. Epub 2023 Oct 27. PMID 37897121
- [Background] Magyar CL, Murdock DR, Burrage LC, Dai H, Lalani SR, Lewis RA, Lin Y, Astudillo MF, Rosenfeld JA, Tran AA, Gibson JB; Undiagnosed Diseases Network; Bacino CA, Lee BH, Chao HT. PRUNE1 c.933G>A synonymous variant induces exon 7 skipping, disrupts the DHHA2 domain, and leads to an atypical NMIHBA syndrome presentation: Case report and review of the literature. Am J Med Genet A. 2022 Jun;188(6):1868-1874. doi: 10.1002/ajmg.a.62704. Epub 2022 Feb 23. PMID 35194938
- [Background] Handoko M, Emrick LT, Rosenfeld JA, Wang X, Tran AA, Turner A, Belmont JW; Undiagnosed Diseases Network; Lee BH, Bacino CA, Chao HT. Recurrent mosaic MTOR c.5930C > T (p.Thr1977Ile) variant causing megalencephaly, asymmetric polymicrogyria, and cutaneous pigmentary mosaicism: Case report and review of the literature. Am J Med Genet A. 2019 Mar;179(3):475-479. doi: 10.1002/ajmg.a.61007. Epub 2018 Dec 19. PMID 30569621
- [Background] Silverman EK, Allard P, Loscalzo J, Mulvihill JJ, Korrick SA; Undiagnosed Diseases Network. Reported environmental exposures are inversely associated with obtaining a genetic diagnosis in the Undiagnosed Diseases Network. Am J Med Genet A. 2019 Jun;179(6):958-965. doi: 10.1002/ajmg.a.61132. Epub 2019 Mar 23. PMID 30903737
- [Background] Macnamara EF, Loydpierson A, Latour YL, D'Souza P, Murphy J, Wolfe L, Estwick T, Johnston JM, Yang J; Undiagnosed Diseases Network; Acosta MT, Lee PR, Pierson TM, Soldatos A, Toro C, Markello T, Adams DR, Gahl WA, Yousef M, Tifft CJ. Risks and benefits of anesthesia for combined pediatric procedures in the NIH undiagnosed diseases program. Mol Genet Metab. 2023 Nov;140(3):107707. doi: 10.1016/j.ymgme.2023.107707. Epub 2023 Oct 10. PMID 37883914
- [Background] Kumble S, Levy AM, Punetha J, Gao H, Ah Mew N, Anyane-Yeboa K, Benke PJ, Berger SM, Bjerglund L, Campos-Xavier B, Ciliberto M, Cohen JS, Comi AM, Curry C, Damaj L, Denomme-Pichon AS, Emrick L, Faivre L, Fasano MB, Fievet A, Finkel RS, Garcia-Minaur S, Gerard A, Gomez-Puertas P, Guillen Sacoto MJ, Hoffman TL, Howard L, Iglesias AD, Izumi K, Larson A, Leiber A, Lozano R, Marcos-Alcalde I, Mintz CS, Mullegama SV, Moller RS, Odent S, Oppermann H, Ostergaard E, Pacio-Miguez M, Palomares-Bralo M, Parikh S, Paulson AM, Platzer K, Posey JE, Potocki L, Revah-Politi A, Rio M, Ritter AL, Robinson S, Rosenfeld JA, Santos-Simarro F, Sousa SB; Undiagnosed Diseases Network; Weber M, Xie Y, Chung WK, Brown NJ, Tumer Z. The clinical and molecular spectrum of QRICH1 associated neurodevelopmental disorder. Hum Mutat. 2022 Feb;43(2):266-282. doi: 10.1002/humu.24308. Epub 2021 Dec 11. PMID 34859529
- [Background] Tinker RJ, Bastarache L, Ezell K, Kobren SN, Esteves C, Rosenfeld JA, Macnamara EF, Hamid R, Cogan JD, Rinker D, Mukharjee S, Glass I, Dipple K, Phillips JA 3rd; Undiagnosed Diseases Network. The contribution of mosaicism to genetic diseases and de novo pathogenic variants. Am J Med Genet A. 2023 Oct;191(10):2482-2492. doi: 10.1002/ajmg.a.63309. Epub 2023 May 29. PMID 37246601
- [Background] Gahl WA, Wise AL, Ashley EA. The Undiagnosed Diseases Network of the National Institutes of Health: A National Extension. JAMA. 2015 Nov 3;314(17):1797-8. doi: 10.1001/jama.2015.12249. No abstract available. PMID 26375289
- [Background] Schymick J, Leahy P, Cowan T, Ruzhnikov MRZ, Gates R, Fernandez L, Pramanik G; Undiagnosed Diseases Network; Yarlagadda V, Wheeler M, Bernstein JA, Enns GM, Lee C. Variable clinical severity in TANGO2 deficiency: Case series and literature review. Am J Med Genet A. 2022 Feb;188(2):473-487. doi: 10.1002/ajmg.a.62543. Epub 2021 Oct 19. PMID 34668327
- [Derived] Keehan L, Carter JN, Kravets E, Wheeler MT, Bernstein JA, Maselli RA, Sampson JB, Bachir S. RAPSN-Associated Congenital Myasthenic Syndrome due to Biallelic Single Nucleotide Variants at the Same Position. Case Rep Genet. 2025 Oct 20;2025:1882021. doi: 10.1155/crig/1882021. eCollection 2025. PMID 41158980
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-HG-0130.html
- See also: https://undiagnosed.hms.harvard.edu — https://undiagnosed.hms.harvard.edu